### Janssen Research & Development

# Statistical Analysis Plan (Week 96 Analysis)

A Phase 3, randomized, active-controlled, open-label study to evaluate switching to a darunavir/cobicistat/emtricitabine/tenofovir alafenamide (D/C/F/TAF) once-daily single-tablet regimen versus continuing the current regimen consisting of a boosted protease inhibitor (bPI) combined with emtricitabine/tenofovir disoproxil fumarate (FTC/TDF) in virologically-suppressed, human immunodeficiency virus type 1 (HIV-1) infected subjects

### Protocol TMC114IFD3013; Phase 3

D/C/F/TAF (darunavir/cobicistat/emtricitabine/tenofovir alafenamide)

**Status:** Final

**Date:** 28 March 2018

**Prepared by:** Janssen Research & Development, a division of Janssen Pharmaceutica NV

**Document No.:** EDMS-ERI-153965642

Compliance: The study described in this report was performed according to the principles of Good Clinical Practice (GCP).

#### **Confidentiality Statement**

The information in this document contains trade secrets and commercial information that are privileged or confidential and may not be disclosed unless such disclosure is required by applicable law or regulations. In any event, persons to whom the information is disclosed must be informed that the information is privileged or confidential and may not be further disclosed by them. These restrictions on disclosure will apply equally to all future information supplied to you that is indicated as privileged or confidential.

# **TABLE OF CONTENTS**

| TABL | LE OF CONTENTS | 2 |
|---|---|---|
| ABBI | REVIATIONS | 4 |
| 1. | INTRODUCTION | 5 |
| 1.<br>1.1. | Trial Objectives | |
| 1.1. | Trial Design | |
| 1.3. | Statistical Hypotheses for Trial Objectives | |
| 1.4. | Sample Size Justification | |
| 1.5. | Randomization and Blinding | |
| 2. | GENERAL ANALYSIS DEFINITIONS | 8 |
| 2.4. | Treatment Arms | 8 |
| 2.5. | Visit Windows | |
| 2.5.1. | | |
| 2.5.2 | | |
| 2.6. | Analysis Sets | |
| 2.6.1. | | |
| 2.6.2 | • | |
| 2.6.3 | | |
| 2.7. | Definition of Subgroups | |
| 2.7.1. | | |
| 2.7.2. | | |
| 2.8. | Re-classification of Stratification Factor for Purpose of Analysis | |
| 2.9. | Reference | 13 |
| _ | OUR LEGT INFORMATION | 40 |
| <b>3.</b> 3.4. | SUBJECT INFORMATION | |
| 3.4.<br>3.5. | Demographics and Baseline Characteristics | |
| 3.6. | Treatment Adherence | |
| 3.0.<br>3.7. | Extent of Exposure | |
| 3.8. | Protocol Deviations | |
| 3.9. | Concomitant Medications | |
| 3.9. | Conconnitant Medications | 14 |
| | EFFICACY | |
| 4.4. | Analysis Specifications | |
| 4.4.1. | | |
| 4.4.2. | | |
| 4.4.2. | 5 · | |
| 4.5. | Primary Efficacy Endpoint | - |
| 4.5.1. | | |
| 4.5.2. | · <b>/</b> · | |
| 4.6. | Major Secondary Efficacy Endpoints | |
| 4.6.1. | | |
| 4.6.2 | • | |
| 4.7. | Resistance Determinations | |
| 4.7.1. | 71 | |
| 4.7.2. | 2. Phenotype | 20 |
| 5. | SAFETY | <mark>21</mark> |
| 5.4. | Adverse Events | |
| 5.4.1. | . Definitions | <mark>21</mark> |

### D/C/F/TAF

(darunavir/cobicistat/emtricitabine/tenofovir alafenamide)

| | Statistical Analysis Plan TMC114IFD3013 (Week | 96) |
|---|---|---|
| 5.4.2. Analysis Methods | | 22 |
| 5.5. Clinical Laboratory Tests | | 23 |
| 5.5.2. Analysis Methods | | 24 |
| | on | |
| 5.5.3.1. Serum Creatinine and Cystatin C | S | 24 |
| | n Findings | |
| REFERENCES | | 30 |
| ATTACHMENTS | | 31 |
| ATTACHMENT 1: PREDEFINED MAJOR P CURRENT LIST | ROTOCOL DEVIATIONS-BASED ON THE | 32 |
| ATTACHMENT 2 | | 36 |
| ATTACHMENT 3 | | 46 |
| ATTACHMENT 4 | | 49 |

#### **ABBREVIATIONS**

AΕ adverse event

alanine aminotransferase ALT

ARV antiretroviral

**AST** aspartate aminotransferase

atazanavir ATV

bone investigation substudy BIS **BMD** bone mineral density BMI body mass index

boosted protease inhibitor bPI confidence interval CI

CKD-EPI Chronic Kidney Disease Epidemiology Collaboration

COBI cobicistat

Division of AIDS **DAIDS** 

D/C/F/TAF darunavir/cobicistat/emtricitabine/tenofovir alafenamide

**DMC** Data Monitoring Committee DPS **Data Presentation Specifications** 

DRV darunavir

estimated glomerular filtration rate eGFR eGFR for creatinine clearance eGFRcr eGFR for cystatin C clearance eGFRcyst early study treatment discontinuation **ESTD** Food and Drug Administration **FDA** 

FDC fixed-dose combination

emtricitabine FTC GSI Gilead Sciences, Inc.

HIV-1 human immunodeficiency virus type 1

ITT Intent-to-Treat LPV lopinavir

MedDRA Medical Dictionary for Regulatory Activities **NCEP** National cholesterol education program

RAM resistance-associated mutation

RNA ribonucleic acid

rtv ritonavir

serious adverse event SAE Statistical Analysis Plan SAP tenofovir alafenamide TAF TDF

tenofovir disoproxil fumarate

TFV tenofovir VL viral load

#### 1. INTRODUCTION

This Statistical Analysis Plan (SAP) describes the W96 analysis that will be performed after the last subject enrolled in the open-label extension phase completes the Week 96 visit, or prematurely discontinues from the study. The final analysis will be described in a separate SAP.

### 1.1. Trial Objectives

The <u>primary objective</u> of this study was to demonstrate noninferiority in efficacy of a D/C/F/TAF oncedaily single-tablet regimen relative to continuing the current bPI combined with FTC/TDF in virologically-suppressed (HIV-1 RNA <50 copies/mL) HIV-1 infected subjects, in regard to the proportion of virologic rebounders (defined as having confirmed HIV-1 RNA  $\ge$ 50 copies/mL through Week 48, or in case of early discontinuation a last single viral load of HIV-1 RNA  $\ge$ 50 copies/mL) with a maximum allowable difference of 4%.

The secondary objectives of this study were:

- To evaluate superiority of switching to a D/C/F/TAF once-daily single-tablet regimen versus continuing the current bPI combined with FTC/TDF in regard to the proportion of virologic rebounders through Week 48, in case noninferiority is established;
- To evaluate the proportion of rebounders through Week 48 in the 2 treatment arms;
- To evaluate efficacy as determined by continued suppression of HIV-1 RNA (<20, <50, and <200 HIV-1 RNA copies/mL as defined by the FDA Snapshot analysis and time to loss of virologic response [TLOVR] algorithm) at Weeks 24 and 48 in the 2 treatment arms;
- To evaluate the safety and tolerability of the D/C/F/TAF regimen through 24 and 48 weeks of treatment;
- To evaluate the change from baseline in serum creatinine, eGFR for creatinine clearance (eGFRcr, by Cockcroft-Gault and by Chronic Kidney Disease Epidemiology Collaboration [CKD-EPI]) and eGFR for cystatin C clearance (eGFRcyst, by CKD-EPI) in the 2 treatment arms at Weeks 24 and 48;
- To evaluate the change from baseline in renal biomarkers at Weeks 24 and 48;
- To evaluate immunologic changes (CD4+ cell count) through 24 and 48 weeks of treatment in the 2 treatment arms;
- To evaluate adherence through drug intake (as derived by drug accountability data), and explore correlation with primary efficacy outcome;
- To evaluate resistance in subjects who show virologic rebound through Weeks 24 and 48 in the 2 treatment arms;
- To evaluate the steady-state pharmacokinetics of DRV in the D/C/F/TAF arm.

<u>Secondary objectives in a bone investigation substudy</u> performed at selected study sites:

- To evaluate the changes from baseline in bone biomarker levels at Weeks 24 and 48;

To evaluate the safety of the 2 treatment arms as determined by the percent change from baseline in spine and hip bone mineral density (BMD) and changes in associated T-score at Weeks 24 and 48.

#### The secondary objectives to be assessed in the study extension:

- To evaluate long-term safety, resistance, and efficacy of the D/C/F/TAF regimen (until Week 96 and beyond).

# 1.2. Trial Design

This is a randomized, active-controlled, open-label, multicenter, Phase 3 study to evaluate the efficacy, safety and tolerability of switching to a D/C/F/TAF once-daily single-tablet regimen compared to continuing the current regimen consisting of a bPI (limited to DRV once daily with rtv or COBI, ATV with rtv or COBI, or LPV with rtv) combined with FTC and TDF (FDC; hereafter referred to as FTC/TDF) in virologically-suppressed (HIV-1 RNA <50 copies/mL), HIV-1 infected adult subjects over a 48-week treatment period.

The aim was to include approximately 1100 subjects in this study. Eligible subjects were to be currently treated with a stable ARV regimen consisting of a bPI (limited to DRV once daily with rtv or COBI, ATV with rtv or COBI, or LPV with rtv) combined with FTC/TDF only, for at least 6 consecutive months preceding the screening visit, and virologically suppressed with at least 1 plasma HIV-1 RNA measurement <50 copies/mL (or HIV-1 RNA undetectable by a local HIV-1 RNA test) occurring between 12 and 2 months prior to screening while being on the stable ARV regimen and have HIV-1 RNA <50 copies/mL at the screening visit. A single viral load elevation of ≥50 copies/mL and <200 HIV-1 RNA copies/mL after previously reaching viral suppression ('blip') within 12 months prior to screening is allowed, provided a subsequent viral load measurement is <50 HIV-1 RNA copies/mL (or HIV-1 RNA undetectable by a local HIV-1 RNA test) prior to screening. A change in pharmacokinetic booster (i.e., rtv or COBI) was allowed provided such a switch occurred no less than 1 month prior to the screening visit. Subjects treated with the combination DRV + COBI + FTC/TDF and having completed the required visits in the Gilead Sciences Inc. (GSI)-sponsored study GS-US-216-0130, and who fulfilled the present protocol criteria, were also given the option to participate in this study.

Prior to or at the baseline visit (Day 1), subjects who met all eligibility criteria were to be randomized in a 2:1 ratio to one of the following 2 treatment arms:

- D/C/F/TAF Arm: Switch to regimen of a single FDC tablet containing DRV 800 mg/ COBI

150 mg/ FTC 200 mg/ TAF 10 mg (D/C/F/TAF tablet) once daily, (n = 734);

- Control Arm: Continue current regimen consisting of a bPI (limited to DRV once daily with

rtv or COBI, ATV with rtv or COBI, or LPV with rtv) combined with FTC/TDF

only, (n = 367).

Randomization was stratified by the bPI used at screening.

Subjects from the D/C/F/TAF arm entered in the extension phase once they had completed their Week 48 visit. In addition, subjects in the control arm received the D/C/F/TAF tablet in the extension phase if, according to the investigator, they benefitted from it and if all conditions were fulfilled (which included adequate viral load results). Subjects from the control arm were required to attend a switch visit at Week

52 to receive D/C/F/TAF. All subjects in the extension phase had to attend visits every 12 weeks up to Week 96. As from Week 96, all subjects are offered the possibility to continue D/C/F/TAF treatment, if they wish and if they continue to benefit from it, until D/C/F/TAF becomes commercially available and is reimbursed, or can be accessed through another source in the country where he/she is living, or until the sponsor terminates clinical development. After Week 96, subjects should attend visits every 6 months.

Subjects who prematurely discontinued or changed study treatment during the treatment phase (from Day 1 to Week 48) or during the extension phase (only between Week 48 and 96) were required to complete the early study treatment discontinuation (ESTD) visit assessments within 72 hours of stopping/changing study treatment.

In addition, a 30-day follow-up (FU) visit was required for any subject who had an ongoing AE or serious adverse event (SAE) at the time of his/her last study visit (unless consent is withdrawn).

The study had a screening period of approximately 30 days starting from the signature of the informed consent form (ICF), a controlled treatment period of 48 weeks, an extension phase up to Week 96 and will have an optional extension beyond Week 96. A 30-day FU visit may take place as described above. A diagram of the study design is provided in Figure 1.

Figure 1: Schematic Overview of the Study

| Baseline<br>(Day 1) | | | ek 48 Wanalysis | eek 96 or<br>beyond |
|---|---|---|---|---|
| Screening | Treatment | t phase | Extension phase | Follow-<br>up |
| ≤30 days prior to<br>baseline | Treatment arm 2 (Control): | | D/C/F/TAF | ESTD<br>and/or<br>30-day<br>FU visit |

A planned Week 24 interim analysis was performed after the last subject completed 24 weeks on study, or prematurely discontinued from the study. The analysis was done mainly to evaluate the safety and tolerability of D/C/F/TAF. However, efficacy of the 2 treatment arms was also assessed and the results were shared with the DMC. The primary Week 48 analysis was performed after the last subject enrolled in the D/C/F/TAF arm reached Week 48 or the last subject enrolled in the control arm completed the Week 52 visit (whichever comes last), or prematurely discontinued from the study. The Week 96 analysis will be performed after the last subject completes 96 weeks on study, or prematurely discontinues from the study. The final analysis will be performed after all subjects have completed the extension phase (and the 30-day FU visit, if applicable).

The efficacy, as well as safety and tolerability, of the enrolled subjects and treatment regimens were monitored by an external DMC until Week 24 analysis.

### 1.3. Statistical Hypotheses for Trial Objectives

No formal statistical hypothesis is to be tested in the Week 96 analysis.

### 1.4. Sample Size Justification

A sample size of 1100 subjects yields 89% power. It was assumed that both treatment arms have a rebound rate of 4% (confirmed HIV-1 RNA  $\geq$ 50 copies/mL up to, and including the upper bound of the Week 48 window or have discontinued prematurely, irrespective of reason, having the last available HIV-1 RNA  $\geq$ 50 copies/mL), that the noninferiority margin is 4%, and that the significance level of the test is at a 1-sided, 0.025 level.

For the bone investigation substudy, with 300 subjects (200 in the D/C/F/TAF treatment arm versus 100 in the control arm) and assuming an inter-subject variability of 4%, there is approximately 98% power to detect a 2% difference between the D/C/F/TAF treatment arm and the control arm in percent change from baseline in BMD at the lumbar spine. Other power calculations are presented below.

BMD at the Lumbar Spine, Power Calculations

| | Mean % Change from | Common Standard | Power |
|-------|--------------------|-----------------|-------|
| | Baseline | Deviation (%) | |
| | 2 | 3.5 | >99% |
| N=300 | 2 | 4 | 98% |
| | 3 | 3.5 | >99% |
| | 3 | 4 | >99% |

### 1.5. Randomization and Blinding

#### Randomization

Central randomization was implemented in this study. Subjects were randomized in a 2:1 ratio to the investigational treatment arm (switch to D/C/F/TAF tablet), or the active control arm (maintain current regimen consisting of a bPI combined with FTC/TDF only). Randomization was stratified by the bPI used at screening (DRV with rtv or COBI, ATV with rtv or COBI, LPV with rtv). Randomization was based on a computer-generated schedule, constructed via random permuted blocks to ensure balance across treatment arms in each stratum of the stratification factors, and prepared before the start of the study by or under the supervision of the sponsor.

#### Blinding

As this is an open-label study, blinding procedures are not applicable.

#### 2. GENERAL ANALYSIS DEFINITIONS

### 2.4. Treatment Arms

Following notations for the treatment arms in extension will be used:

- **Initial switch to D/C/F/TAF**: subjects who received D/C/F/TAF treatment at baseline of the treatment phase (initial switchers)
- **Late switch to D/C/F/TAF**: subjects who continued on their bPI treatment for 52 weeks and who switched to D/C/F/TAF treatment in the extension (late switchers)

#### 2.5. Visit Windows

### 2.5.1. Trial Phases

Phases will be constructed for each subject as follows for adverse events, concomitant therapies, and for the determination of the worst-case/toxicity/change in the cross-tabulations.

| Trial phase | Start date | End date |
|---|---|---|
| Screening | Minimum of Date of signing the informed consent and Date of the screening visit | 1 day before start of treatment |
| Comparative<br>Treatment<br>Phase | Date of the first intake (after randomization) | <ul> <li>For initial D/C/F/TAF subjects, in order of priority: <ul> <li>Week 48 visit date; if missing then</li> <li>Projected Week 48 visit date, where projected Week 48 visit date = baseline visit date + (7 *48)</li> </ul> </li> </ul> |
| | | For late switchers: |
| | | Date of first D/C/F/TAF intake-1 day |
| | | In case of withdrawal use: |
| | | <ul> <li>Minimum(last intake date of study drug, study withdrawal date) + 2 days</li> </ul> |
| Extended<br>Treatment<br>Phase<br>(Extension) | Last Date of Comparative<br>Treatment Phase +1 day | <ul> <li>Week 96 visit date; if missing then</li> <li>Projected Week 96 visit date, where projected Week 96 visit date = baseline visit date + (7 *96)</li> </ul> |
| | | <ul><li>In case of withdrawal use:</li><li>Minimum (last intake date of study drug, study withdrawal date) + 2 days</li></ul> |
| Follow-up | End of last treatment phase +1 day | Trial termination date for all groups (date of last contact) |

Data up to each subject's Week 96 visit are in scope for this analysis, DXA data (DP domain) up to Week 96 visit+28 days, and if applicable, any (confirmatory) viral load or genotype/phenotype results immediately subsequent to Week 96 (up to 6 weeks).

### 2.5.2. Analysis Time points

All visits/assessments will be allocated to the following time points as per the table below, based on the number of days in the study, calculated as "assessment date – start date of comparative treatment phase + 1 day" for Comparative Treatment/Extended treatment and Follow-up phase.

The following time intervals will be used for reporting of efficacy as well as safety data:

| Phase | Visit | Target day | Analysis time point | Time interval (days) |
|---|---|---|---|---|
| Screening | 1 | -∞ | Screening | < Day 0 |
| Comparative | 2 | 1 | Baseline <sup>a</sup> | ≤Day 1 |
| Treatment | 3 | 15 | Week 2 | Day 2 – Day 21 |
| Phase | 4 | 29 | Week 4 | Day 22 – Day 42 |
| | 5 | 57 | Week 8 | Day 43 – Day 70 |
| | 6 | 85 | Week 12 | Day 71 – Day 126 |
| | 7 | 169 | Week 24 | Day 127 – Day 210 |
| | 8 | 253 | Week 36 | Day 211 – Day 294 |
| | 9 | 337 | Week 48 <sup>b</sup> | Day 295 – Day 378 |
| Extended treatment | 10 | 421 | Week 60 (Week 12) | Day 379 – Day 462 |
| phase (Extension) | 11 | 505 | Week 72 (Week 24) | Day 463 – Day 546 |
| | 12 | 589 | Week 84 (Week 36) | Day 547 – Day 630 |
| | 13 | 673 | Week 96 <sup>c</sup> (Week 48) | Day 631 – Day 714 |
| Follow-up | 14 | 31 | Follow-up | Day 1 onwards |

<sup>&</sup>lt;sup>a</sup> Only the record closest to target day 1 will be allocated to analysis time point 'Baseline', all records prior to day 1 are assigned to 'Screening'.

Note, for Initial Switchers to D/C/F/TAF, period "Baseline-Week 96" will include visits from Comparative treatment phase and Extended treatment phase.

Unless specified otherwise, if two visits fall within the same interval, the one closest to the target day will be used for the analysis displays and graphics in order to have only one evaluation per subject per analysis time point. However, all data will be presented in the listings. If distances of both visits to the target day are equal, the visit latest in time will be used. If multiple visits that fall within the same analysis window have the same date/time, the one with the highest sequence number will be used.

### 2.6. Analysis Sets

# 2.6.1. Intent-to-Treat Analysis Set

The intent-to-treat (ITT) analysis set includes all the subjects who were randomized and received at least 1 dose of treatment subsequent to randomization in the study. Efficacy data up to the last dose date of the treatment are included. The safety analysis (including all data collected at the 30-day FU visit) is also performed on this analysis set.

### 2.6.2. Per Protocol Analysis Set

An analysis based on the per protocol (PP) population will also be performed to investigate the impact of excluding subjects with major protocol violations and to evaluate the robustness of the analysis results. The PP population will include all subjects who:

For DXA scans a scan up to 28 days post-baseline was used as a baseline scan.

<sup>&</sup>lt;sup>b</sup> DXA scan up to 28 days post-Week 48 was used as the Week 48 scan

<sup>&</sup>lt;sup>c</sup> DXA scan up to 28 days post-Week 96 was used as the Week 96 scan.

- (1) are randomized into the study,
- (2) have received  $\geq 1$  dose of treatment in the study, and
- (3) without any major protocol deviation that is considered to potentially affect efficacy outcomes. Specific details are provided in Attachment 1.

The PP analysis set is the secondary analysis set for efficacy analysis. The per protocol (PP) set is defined as the ITT analysis set minus subjects with major protocol violations as listed in Attachment 1

# 2.6.3. Bone Investigation Substudy Analysis Set

The bone investigation substudy (BIS) analysis set includes all subjects in the ITT set and having at least one post-baseline value either in biomarker or in BMD data. The bone investigation analysis will be performed on this analysis set.

### 2.7. Definition of Subgroups

### 2.7.1. Subgroups for Efficacy Analyses

- Adherence based on D/C/F/TAF (i.e., from reference) drug accountability (>95%: adherent, \( \leq 95\)%: non-adherent, missing/unknown)
- Reference viral load
  - o For Initial D/C/F/TAF group the screening and baseline viral load
    - <50; if all screening and baseline viral load values are below 50 copies/mL</p>
    - ≥50; if at least one viral load value during screening or baseline ≥50 copies/mL)
  - o For Late Switch group, the reference viral load
    - <50 copies/mL</p>
    - ≥50 copies/mL
- CD4+ count at reference (<200,  $\ge 200$  [ $200 \le x < 350$ ,  $350 \le x \le 500$ , >500] cells/mm<sup>3</sup>)
- Race (American Indian or Alaska Native, Asian, Black or African American, White, Native Hawaiian or other Pacific Islander, Other, non-Black or African American)
- Ethnicity (Hispanic or Latino, non-Hispanic or Latino)
- Gender (Female, Male)
- Age group ( $\leq$ 50, >50 years)
- Region (Europe, North America)
- Re-classified bPI at screening (see section 2.5):
  - o DRV once daily with rtv or COBI; ATV with rtv or COBI; LPV with rtv
  - o ATV with rtv or COBI, or LPV with rtv
  - o DRV with rtv; DRV with COBI
- Booster at screening (ritonavir or cobicistat)
- Number of previous ARVs used (3, 4, 5, 6, 7, >7) and previous PI, N(t)RTI or NNRTI used (0, 1, 2, 3, 4, >4)

- Previous ARV failure and previous PI, N(t)RTI or NNRTI failure  $(0, \ge 1)$
- WHO Clinical Staging of HIV/AIDS
- Viral blip (see section 4.6.1) during first 48 weeks:
  - Yes, if subject experience at least 1 viral blip during the first 48 weeks of the study
  - No, otherwise
- For the Late Switch group only:
  - Protocol-defined virologic rebound during first 48 weeks
    - Yes, if subject experience a protocol-defined virologic rebound during the first
       48 weeks of the study
    - No, otherwise

### 2.7.2. Subgroups for Safety Analyses

- Race (American Indian or Alaska Native, Asian, Black or African American, White, Native Hawaiian or other Pacific Islander, Other, non-Black or African American)
- Ethnicity (Hispanic or Latino, non-Hispanic or Latino)
- Gender (Female, Male)
- Age group ( $\leq$ 50, >50 years)
- Region (Europe, North America)
- Re-classified bPI at screening:
  - o DRV once daily with rtv or COBI; ATV with rtv or COBI; LPV with rtv
  - o ATV with rtv or COBI, or LPV with rtv
  - o DRV with rtv; DRV with COBI
- Booster at screening (ritonavir or cobicistat)
- Reference eGFR<sub>CG</sub> ( $<70, \ge 70 \text{ mL/min}$ )
- WHO Clinical Staging of HIV/AIDS

Subgroups for Bone Investigation Analyses:

- o bPI at screening
- o Race (American Indian or Alaska Native, Asian, Black or African American, White, Native Hawaiian or other Pacific Islander, Other, Non Black)
- Gender
- o Reference BMI ((underweight ( $<18.5 \text{ kg/m}^2$ ), normal range ( $18.5 \text{ to } <25.0 \text{ kg/m}^2$ ), overweight ( $\ge 25.0 \text{ kg/m}^2$ ) and obese ( $\ge 30.0 \text{ kg/m}^2$ ))

- o Age group ( $\leq 50$ ,  $\geq 50$  years)
- Current smoking status (yes/no)

### 2.8. Re-classification of Stratification Factor for Purpose of Analysis

For the purpose of analysis the stratification factor (bPI) was re-classified based on the value from the history of ARV therapy data at screening.

The re-classified stratification factor is used for analysis..

#### 2.9. Reference

For Initial D/C/F/TAF group, reference is the comparative treatment phase baseline as in Week 48 analysis. For the late switch group two references will be used: (1) comparative treatment baseline will be used as reference for the period up to the switch; (2) the last value prior to the switch will be used as reference for the extended treatment phase.

#### 3. SUBJECT INFORMATION

### 3.4. Demographics and Baseline Characteristics

These parameters will not be included in this analysis, because no new subjects were recruited since the Week 48 analysis.

#### 3.5. Disposition Information

A tabulation of the total number (with percentages) of subjects screened, randomized and not treated, randomized and treated in extended treatment phase will be provided.

Tabulation per treatment arm and overall of the number of subjects who have completed the treatment/extended treatment phase, who are ongoing, and who have discontinued the trial before Week 96 visit, with the reason for discontinuation will be provided.

A Kaplan-Meier graph for the time to Discontinuation (any reason) will be included.

#### 3.6. Treatment Adherence

Treatment adherence based on drug accountability will be summarized by means of descriptive statistics and frequency tabulations. Cumulative treatment adherence will be calculated from baseline through Week 96 for the Initial Switch to D/C/F/TAF arm; from baseline to the switch, and again from the switch to Week 96 for the Late Switch to D/C/F/TAF arm. Cumulative treatment adherence will be determined (derivation i).

The following parameters are derived:

Amount to be taken through switch/Week 96 = (number of days since start of treatment/switch  $\times$  number of tablets to be taken per day).

Number of days since start of treatmentswitch is based on (whichever comes sooner):

- <u>last study medication intake</u> (if available) or, in case subject discontinued and last study medication intake is missing, the last visit date prior to withdrawal will be used.
- Switch/Week 96 visit date

In addition (derivation ii), the cumulative treatment adherence up to time point where not more than one bottle is missing, or if available, up to switch/Week 96, whichever comes sooner, will be calculated.

**Actual amount taken** = (number of tablets dispensed – number of tablets returned), summed over time points up to the time point of interest.

**Level of adherence** = (actual amount taken / amount to be taken)  $\times$  100%

Treatment adherence is defined as:

- adherent: the level of adherence is >95%,
- non-adherent: the level of adherence is  $\leq 95\%$ .

Additionally, following categories of level of adherence will be defined:

- >95%
- [80%; 95%]
- [65%; 80%]
- [50%; 65%]
- $\le 50\%$

Interruptions (for AEs) are not to be taken into account for the calculation of adherence, i.e. they will not be subtracted from the amount to be taken.

# 3.7. Extent of Exposure

Descriptive statistics will be tabulated for the duration of treatment of both treatment groups, in weeks, during the respective active treatment phases, as of reference, up to the Week 96 visit, or in case of early discontinuation, last study medication intake. In addition, subject-years of exposure will be shown, derived as mean of treatment duration ((in weeks)  $\times$  N)  $\times$  7 / 365.25.

Treatment duration (in weeks) is derived as follows:

```
(End of phase - reference + 1) / 7
```

Treatment interruptions will not be taken into account for the above definition.

#### 3.8. Protocol Deviations

All major protocol deviations will be tabulated and listed by treatment arm and overall. The proportion of subjects with one or more major protocol deviation that led to exclusion from the per protocol analysis set (Attachment 1) will also be tabulated.

### 3.9. Concomitant Medications

Concomitant medications are defined as any therapy used on or after the same day as the first dose of study agent, including those that started before and continue on after the first dose of study agent. Combination drugs are split up into their respective compounds. When counting the number of ARVs at a specific time point or during a specific time period, the separate compounds of these combination drugs are counted

Concomitant therapies will be grouped as follows, using a list of dictionary derived terms provided as metadata. These groups will be tabulated (n, %) per treatment group and analysis phase:

- lipid lowering drugs
- antidiabetic drugs
- antihypertensive drugs
- drugs for cardiovascular disease
- antiosteoporotic drugs

#### 4. EFFICACY

### 4.4. Analysis Specifications

### 4.4.1. Level of Significance

No formal statistical tests will be calculated. All results will be descriptive.

### 4.4.2. Data Handling Rules

Plasma viral load levels will be measured using the ROCHE COBAS® AmpliPrep/COBAS® Taqman® HIV-1 Test, v2.0 assay, which will be conducted by the central laboratory.

Imputation of left censored HIV-1 RNA values: viral load results recorded as "< 20 HIV-1 RNA copies/mL detected" and "< 20 HIV-1 RNA copies/mL not detected" will be scored at 19.

CD4+ cell count and HIV-1 RNA data collected on treatment (up to the last dose date of study drug) will be used in the analysis.

### 4.4.2.1. Data Handling for Late Switchers

Except for analyses by analysis time point or change from baseline, data (i.e., Protocol-defined virologic rebound through Week96, Snapshot at Week 96, TLOVR and Resistance analyses) from the Late Switch to D/C/F/TAF group will be presented in tables and figures from the reference onwards to Week 96.

### 4.5. Primary Efficacy Endpoint

#### 4.5.1. Definition

The primary efficacy endpoint of this study was the proportion of subjects with protocol-defined virologic rebound cumulatively through 48 weeks. Thus, the analysis of this endpoint is not described in the Week 96 SAP.

### 4.5.2. Analysis Methods

Not applicable.

#### 4.6. Major Secondary Efficacy Endpoints

- The proportion of subjects with protocol-defined virologic rebound based on the HIV-1 RNA ≥50, ≥20 and ≥200 copies/mL threshold through 96 weeks;

- The proportion of subjects with virologic response and failure based on the 20, 50 and 200 copies/mL threshold at Week 96, as defined by the FDA Snapshot approach (4.6.1);
- The proportion of subjects with virologic response and failure based on the 20, 50 and 200 copies/mL at Week 96, as defined by the TLOVR algorithm (4.6.1);
- Time to virologic rebound up to Week 96
- The change from reference in CD4+ cell count
- The proportion of subjects with viral blip based on the HIV-1 RNA ≥50 and ≥200 copies/mL threshold through 96 weeks

#### 4.6.1. Definitions

#### Virologic Rebound

Virologic rebound is defined as:

- subjects who show confirmed HIV-1 RNA ≥50/20/200 copies/mL from the reference up to, and including Week 96,
- subjects who discontinued prematurely (irrespective of reason) for which the last available (single) HIV-1 RNA value on treatment was ≥50/20/200 copies/mL.
- any subject with last available on-treatment HIV-1 RNA ≥50/20/200 copies/mL at the study cutoff of Week 96 (i.e., any last viral load [re]test having occurred no later than 6 weeks after Week 96)

All other situations are considered non-rebounders.

### Snapshot approach (applying 20/50/200 copies/mL as threshold)

The Snapshot approach will classify subjects into 3 outcome categories: "virologic success", "virologic failure" and "No viral load data". Several subcategories of the outcome will also be presented in the analysis and are shown below. The categories below are mutually exclusive such that a subject will be included in one (sub)category. If a subject discontinues in the time window but also has an HIV-RNA value in the time window then the viral load data will be used to classify the subject's category.

- Virologic success:
  - Last available HIV RNA <20/50/200 copies/mL in the Week 96 visit window (Week 90-102)
- Virologic failure:
  - Last available HIV RNA ≥20/50/200 copies/mL in the Week 96 visit window (Week 90-102)
  - Virologic failure leading to discontinuation

- o Discontinued due to other reason (i.e. other than AE/death or virologic failure) and last available HIV-RNA ≥20/50/200 copies/mL
- No viral load data in the Week 96 visit window
  - Discontinued due to AE/death (subjects will be classified in this category if discontinued prior to Week 96 window regardless of HIV-RNA level)
  - Discontinued due to other reason (i.e. other than AE/death or virologic failure) and the last available HIV RNA <20/50/200 copies/mL (or missing)</li>
  - o Missing data during the Week 96 visit window but on study

The following threshold criteria are considered:

- <20: HIV RNA below 20 copies/mL (target not detected or target detected)
- <50: HIV RNA below 50 copies/mL
- <200: HIV-RNA below 200 copies/mL

#### **Imputations for missing values**

The following imputation method is used to calculate **virologic response** at a given time point:

- observed case: subjects with a missing value are disregarded in the analysis for that time point.
- <u>TLOVR</u>: responders/non-responders are defined according to the FDA Time To Loss Of Virologic Response algorithm; a subject is considered a responder at a given time point if the applicable HIV-RNA criterion is fulfilled at that time point and at the subsequent time point; a subject is considered a confirmed non-responder at a time point in the following situations in order of precedence:
  - o the subject (permanently) discontinued at that time point or before
  - o the subject shows a 'rebound' HIV-RNA value (≥threshold copies/mL) at that time point and the subsequent time point;
  - o the subject shows a confirmed rebound at an earlier time point (irrespective of resuppression of viral load)
  - o intermittently missing values are considered as response if the immediately preceding and following visits demonstrated response; in case the subject had not reached the next visit yet, no imputation is performed for the missing time points, unless the subject had discontinued the trial.
  - Remark: in case multiple virologic response observations are available within the same time window, all observations are used to determine TLOVR-imputed response for that time window. In case the subject has not reached the next visit yet, this subject is left out of the analysis for the missing time points.

In addition, TLOVR outcome table at Week 96 will be presented.

<u>Time to rebound:</u> The time (in weeks) calculated from reference until the first rebound time point (time point before confirmation of rebound) up to Week 96 visit. Subjects never losing the response up to Week 96 visit will be censored at the end of the extended treatment phase.

<u>Immunologic response:</u> The change from reference in CD4+ count and CD4% at a given time point is defined as: (CD4+/CD4% at a given time point - reference CD4+/CD4%).

Subjects who discontinue will have their CD4 values after discontinuation imputed with their reference value, thus resulting in a 0 change (NC=F). Other (intermittent) missing values will be imputed using last observation carried forward (LOCF). Apart from imputed, observed data will also be presented.

For cases where <u>no observation is available at the baseline date</u>, the last available screening value will be taken.

<u>Viral Blip:</u> A viral blip is defined as any HIV-1 RNA value ≥50/200 copies/mL preceded and followed by HIV-1 RNA <50/200 copies/mL (a confirmed rebound does not constitute a Blip). All HIV-1 RNA viral load data from the reference point to lower limit of the Week 96 window will be used to classify Viral Blip.

### 4.6.2. Analysis Methods

#### Protocol-defined virologic rebound, Snapshot and TLOVR approach

Tabulations (numbers and proportions) per time point will be provided for the Snapshot outcomes (success, failure, no data within window). Tabulations (numbers and proportions) will also be provided for the categorical parameters (virologic rebounders and TLOVR), through Week 96. The exact 2-sided 95% CIs around in each treatment group will be calculated by the Clopper-Pearson method for Protocoldefined virologic rebound, Snapshot virologic success and virologic failure, and TLOVR response Bar charts will be presented for virologic rebounders and Snapshot outcomes.

#### Time to virologic rebound

Time to virologic rebound will be graphically presented by means of Kaplan-Meier curves and a Cox proportional hazards model will be fit separately for each treatment group. Terms included in the model for the initial D/C/F/TAF group will be bPI at screening, and any pre-dose (screening phase) viral load ≥50 copies/mL (Yes/No). Terms in the model for the Late Switch group will be bPI at screening and any pre-D/C/F/TAF dose viral load ≥50 copies/mL (Yes/No).

#### **Immunologic Change**

Descriptive statistics (n, mean (se), median, and ranges) per time point will be provided for the continuous parameters, CD4 cell count actual values and change from reference. CIs for the means and mean changes will be calculated. The changes from reference (NC=F) of the two treatment arms and the 95% CIs at Week 96 will be constructed using ANCOVA separately for each treatment group, including term for bPI at screening and reference CD4+ value as a covariate. A sensitivity analysis using Mixed-effects model for repeated measures (MMRM) approach will also be performed separately for each treatment. The model will include change from reference as a response variable (observed case), terms for bPI at screening, visit, and the corresponding reference value as a covariate. An unstructured covariance matrix will be used to model the correlation among repeated measurements.

Cross-tabulations of Week 96 CD4 cell count versus reference will be provided using the categories:  $< 200, 200 \le x < 350, 350 \le x \le 500, >500 \text{ cells/mm}^3$ 

#### Viral Blip

Tabulations (numbers and proportions) of subjects with 0, 1, 2, 3 or more blips will be presented. Further, FDA Snapshot outcome at Week 96 and descriptive statistics of adherence by subjects with rebound, Blip or No Blip will be presented. CMH (nonzero correlation) test will be used for comparison within

treatment group of compliant (>95%), Snapshot success as well as for Snapshot failures. Blips will also be presented graphically.

#### Per Protocol Analysis

The key secondary endpoints will also be analyzed on the per protocol (PP) population. Details on which outputs are included for the PP population will be provided in the Data Presentation Specifications (DPS) document.

#### 4.7. Resistance Determinations

Inclusion of subjects for resistance analysis will be based on the availability of post-baseline genotypic/phenotypic data also described below.

### 4.7.1. Genotype

HIV-1 PR/RT genotype will be assessed by the GenoSureMG<sup>TM</sup> assay. Genotypes were requested on eligible samples with a viral load  $\geq$  400 copies/mL. Results will be shown per PR and RT and time point and will be generated in individual listings. Name and date of mutation lists will be indicated.

The analysis aims to characterize the frequency of post-baseline PR and RT resistance mutations in all subjects with genotype data and in subjects with virologic rebound having genotype data.

A tabulation per treatment group will present the number of patients with a specific mutation or number of patients with at least one PR or RT mutation belonging to a specific mutation list (see below). The analysis assumes a worst case scenario in case of multiple post-baseline sequencing results: if any of a patient's samples shows a mutation, the patient is assumed to have this mutation, even if other samples show wild-type virus.

All analyses will be conducted on the Efficacy ITT population, unless specified otherwise.

#### **Protease mutations**

- IAS-USA<sup>2</sup> Primary PI mutations (n=23)
   D30N, V32I, M46I/L, I47A/V, G48V, I50L/V, I54L/M, Q58E, T74P, L76V, V82A/F/L/S/T, N83D, I84V, N88S, L90M
- IAS-USA<sup>2</sup> Secondary PI mutations (n=52)
   L10C/F/I/R/V, V11I, G16E, K20I/M/R/T/V, L24I, L33I/F/V, E34Q, M36I/L/V, K43T, F53L/Y, I54A/S/T/V, D60E, I62V, L63P, I64L/M/V, H69K/R, A71I/L/T/V, G73A/C/S/T, V77I, V82I, I85V, N88D, L89I/M/V, I93L/M
- IAS-USA<sup>2</sup> DRV resistance-associated mutations (n=11)
   V11I, V32I, L33F, I47V, I50V, I54L/M, T74P, L76V, I84V, L89V

#### **RT** mutations

IAS-USA<sup>2</sup> NRTI resistance-associated mutations (n=22)
 M41L, A62V, K65R/E/N, D67N, 69ins, K70E/R, L74V, V75I, F77L, Y115F, F116Y, Q151M, M184I/V, L210W, T215F/Y, K219E/Q

- IAS-USA<sup>2</sup> NNRTI resistance-associated mutations (n=34)
   V90I, A98G, L100I, K101E/H/P, K103N/S, V106A/I/M, V108I, E138A/G/K/Q/R, V179D/F/L/T, Y181C/I/V, Y188C/H/L, G190A/S, H221Y, P225H, F227C, M230I/L
- IAS-USA<sup>2</sup> Thymidine Analogue Mutations (TAMs) (n=8) M41L, D67N, K70R, L210W, T215Y/F, K219Q/E
- IAS-USA<sup>2</sup> TFV resistance-associated mutations K65R/E/N, K70E
- IAS-USA<sup>2</sup> FTC resistance-associated mutations K65R/E/N, M184I/V

# 4.7.2. Phenotype

Predicted phenotype based GenoSureMG<sup>TM</sup> and in-vitro phenotype data, if applicable, based on PhenoSense<sup>TM</sup> HIV assay, will be presented in individual patient listings per drug and time point. Fold change (FC) in 50% effective concentration (EC50) of ARVs versus wild-type HIV-1 virus will be included in individual listings per drug and time point.

PhenoSense<sup>TM</sup> could additionally be requested to determine the phenotypic drug susceptibility of the virus if resistance-associated mutations to the study drugs were observed. Using the fold change (FC), each drug will be categorized into sensitive/partially sensitive/resistant based on cut-off values.

Number and percentage of genotypic/phenotypic susceptibility (i.e., sensitivity) will be tabulated (numbers and proportions) per class and drug.

When one cut-off value is available, a drug is considered

- Sensitive if the FC is below or equal to the clinical cut-off (CCO) when available or below or equal to the biological cut-off (BCO) otherwise;
- Resistant if the FC is above the clinical or biological cut-off.

When two cut-off values are available, a drug is considered

- Sensitive if the FC is below or equal to the lower cut-off;
- Partially sensitive if the FC is above the lower cut-off and below or equal to the higher cut-off;
- Resistant if the FC is above the higher cut-off.

### BCOs and CCOs for the PhenoSense® GT Phenotyping Assay

| Class | Drug | Generic name | PhenoSense GT <sup>TM</sup> (V7045/V7145) |
|-------|------|---------------|-------------------------------------------|
| NRTI | AZT | Zidovudine | 1.9 |
| | 3TC | Lamivudine | 3.5 |
| | ddI | Didanosine | 1.3 - 2.2 |
| | d4T | Stavudine | 1.7 |
| | ABC | Abacavir | 4.5 – 6.5 |
| | FTC | Emtricitabine | 3.5 |
| | TDF | Tenofovir | 1.4 – 4.0 |
| NNRTI | NVP | Nevirapine | 4.5 |

| | DLV | Delavirdine | 6.2 |
|----|---------------------|-------------------------------------|-------------|
| | EFV | Efavirenz | 3.0 |
| | ETR | Etravirine | 2.9 - 10.0 |
| | RLP | Rilpivirine | 2.0 |
| PI | ATV | Atazanavir | 2.2 |
| | ATV/rtv | Boosted Atazanavir | 5.2 |
| | DRV/rtv | Boosted Darunavir | 10.0 - 90.0 |
| | APV/rtv or fAPV/rtv | Boosted Amprenavir or fosamprenavir | 4.0 - 11.0 |
| | IDV/rtv | Boosted Indinavir | 10.0 |
| | LPV/rtv | Boosted Lopinavir (Kaletra) | 9.0 - 55.0 |
| | NFV | Nelfinavir | 3.6 |
| | RTV | Ritonavir | 2.5 |
| | SQV/rtv | Boosted Saquinavir | 2.3 - 12.0 |
| | TPV/rtv | Boosted Tipranavir | 2.0 - 8.0 |

Clinical cut-offs are shown in bold; cutoffs are based on the PhenosenseGT algorithm version 13

#### 5. SAFETY

For initial switchers, comparative treatment phase (study baseline to Week 48), extended treatment phase (Week 48 to Week 96) as well as combination of both phases (study baseline to Week 96) will be presented in the tables. For late switchers, comparative treatment phase (study baseline up to the switch) and extended treatment phase (from the switch to Week 96) will be presented.

#### 5.4. Adverse Events

#### 5.4.1. Definitions

Reported AE parameters and grades are based on the Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events ("**DAIDS AE grading table**"). All AEs will be coded using MedDRA version 20.0.

### **Events of interest**

The EOIs groups include a broad list of terms to identify potential cases. The list of all preferred terms belonging to each AEOI group is provided in Attachment 2.

Since many of the terms used to identify potential cases are clinically non-specific, only those retrieved cases that upon medical review are specifically suggestive of /compatible with the AEs of special interest will be commented on in the CSR.

Adverse events of interest (AEOI) groups used for the safety analyses are the following:

- Renal AEOI (for PRT)

Subgroups: laboratory related events,

clinical events

- Bone AEOI (for fractures)

Subgroups: Osteomalacia,

Bone Loss/atrophy,

Fracture, possibly osteoporotic, Fracture other, Other Bone Events

- Lipid-related AEOI
- Liver AEOI
- Hyperglycemia AEOI
- Pancreas AEOI
- Severe skin AEOI
- Rash AEOI
- Immune reconstitution inflammatory AEOI
- Coronary artery AEOI
- Ocular AEOI (for posterior uveitis)
- Lipodystrophy AEOI
- Cardiac conduction AEOI

Subgroups: Conduction defects,

Torsade de pointes/QT prolongation

Convulsion AEOI

#### **Adverse Drug Reaction (ADR)**

ADRs will be presented. A list of all ADRs is in the Attachment 3. The medical assessment of the safety data was performed according to a pre-specified algorithm and. In case multiple lists are available (US and EU definitions), ADRs will be tabulated separately per list.

### 5.4.2. Analysis Methods

A summary will be provided for the following treatment-emergent adverse events:

- any adverse events,
- serious adverse events.
- deaths due to AE,
- adverse events by toxicity grade (as well as AEs with toxicity grade at least 2 and AEs with toxicity grades 3 or 4),
- AEs at least possibly related to study medication,
- AEs for which the medication was temporarily/permanently stopped,
- serious adverse events that were at least possibly related to the medication.

Incidences of AEs for above mentioned analyses will also be presented by SOC and preferred term. There will be no formal statistical testing.

Summary of events and incidence tabulations for individual adverse events will be provided for AEOI and also for ADRs.

AIDS defining illness based on WHO clinical staging will be tabulated.

The number and percentage of subjects who experienced fracture events (subgroups Fracture, possibly osteoporotic and Fracture other of the Bone AEOI for fractures) will be summarized by treatment group.

Selected safety endpoints will be explored by subgroups defined in section 2.7.2. Details for subgroup analyses of safety endpoints will be provided in the DPS.

### 5.5. Clinical Laboratory Tests

#### 5.5.1. Definitions

Laboratory parameters of the following lab subcategories will be investigated. The results will be displayed grouping the tests as follows:

- General biochemistry:
  - blood: creatine phosphokinase, alpha-1 acid glycoprotein
  - urine/dipstick: blood, nitrite, leukocyte esterase
- Hematology: hematocrit, hemoglobin, platelet count, red blood cell count (RBC), white blood cell count (WBC), mean corpuscular volume (MCV), mean corpuscular hemoglobin (MCH) and mean corpuscular hemoglobin concentration (MCHC)

Hematology differential counts: basophils, eosinophils, lymphocytes, monocytes, neutrophils (counts and %).

#### Laboratory Events of Interest

- Pancreatic parameters: total amylase, lipase
- Liver related parameters:
  - ALT, AST, alkaline phosphatase (ALP), gamma glutamyl transferase (GGT), bilirubin (all types)
  - Urine/dipstick: bilirubin, urobilinogen
- Lipid parameters: cholesterol, HDL cholesterol (HDL-C) (all types), LDL cholesterol (LDL-C) (all types), TC/HDL, triglycerides; these will be analyzed overall irrespective of fasting status as well as restricted to results from fasting samples separately
- Glucose parameters will be analyzed overall irrespective of fasting status as well as restricted to results from fasting samples separately:
  - blood: glucose
  - urine/dipstick: glucose, ketones
- Renal parameters:
  - blood: total protein, creatinine, blood urea nitrogen, uric acid, phosphorus, potassium, sodium, bicarbonate, chloride, albumin
  - urine/chemistry: creatinine, sodium, phosphate, glucose, urine albumin, urine protein
  - urine/dipstick: glucose, protein

Laboratory toxicities will be derived based on the DAIDS toxicity grading scale (see Protocol).

*Note*: Local lab results will not be used for the analyses.

## 5.5.2. Analysis Methods

Descriptive statistics for the actual values and changes from reference will be provided per time point.

Cross-tabulations of the worst toxicity grades through Week 96 versus reference, and cross-tabulations of the worst toxicity grades at Week 96 versus reference will also be provided if applicable. Subject listings of abnormal laboratory values will be provided.

For lipids and renal parameters, within-treatment arm comparison versus reference at Week 96 will be assessed using Wilcoxon signed-rank test.

Additionally, the following lipid-related abnormalities according to NCEP categories will also be tabulated:

- Triglycerides abnormally high (≥150 mg/dL)
- Total cholesterol abnormally high (≥ 200 mg/dL)
- LDL abnormally high ( $\geq 100 \text{ mg/dL}$ )
- HDL abnormally low (< 40 mg/dL)

#### Hy's Law Criteria

In addition, an analysis will be performed to identify all subjects meeting Hy's law criteria i.e. subjects showing 3-fold or greater elevations above the ULN of ALT or AST and a concomitant elevation of serum total bilirubin to >2xULN, without a concomitant elevated serum ALP (defined as serum alkaline phosphatase activity less than  $2\times$  the upper limit of normal).

# 5.5.3. Creatinine and glomerular filtration

### 5.5.3.1. Serum Creatinine and Cystatin C

Estimated glomerular filtration rate based on the creatinine clearance will be calculated according to the Cockcroft-Gault formula<sup>3</sup> (eGFRcr<sub>CG</sub>) and the CKD-EPI formula (eGFRcr<sub>CKD-EPI</sub>) and eGFR based on cystatin C clearance will be calculated according to the CKD-EPI formula (eGFRcyst<sub>CKD-EPI</sub>).

- eGFRcr according to the Cockcroft-Gault formula (unit: mL/min):

Male:  $(140 - age in years) \times (weight in kg) = eGFRcr_{CG}(mL/min)$ 72 × (serum creatinine in mg/dL)

Statistical Analysis Plan TMC114IFD3013 (Week 96)

Female: 
$$(140 - age in years) \times (weight in kg) \times 0.85 = eGFRer_{CG} (mL/min)$$
  
72 × (serum creatinine in mg/dL)

eGFRcr and eGFRcyst according to the CKD-EPI formula (unit: mL/min/1.73m<sup>2</sup>):

### eGFRcr<sub>CKD-EPI</sub>

Female: 
$$Scr \le 0.7 \text{ mg/dL}$$
 144 x  $(Scr/0.7)^{-0.329}$  x 0.993<sup>age</sup> Scr >0.7 mg/dL 144 x  $(Scr/0.7)^{-1.209}$  x 0.993<sup>age</sup> Male:  $Scr \le 0.9 \text{ mg/dL}$  141 x  $(Scr/0.9)^{-0.411}$  x 0.993<sup>age</sup> Scr >0.9 mg/dL 141 x  $(Scr/0.9)^{-1.209}$  x 0.993<sup>age</sup>

#### eGFRcyst<sub>CKD-EPI</sub>

Scyst 
$$\le 0.8 \text{ mg/L}$$
 133 x (Scyst/0,8)<sup>-0.499</sup> x 0.996<sup>age</sup> [x 0.932 if female]  
Scyst  $> 0.8 \text{ mg/L}$  133 x (Scyst/0,8)<sup>-1.328</sup> x 0.996<sup>age</sup> [x 0.932 if female]

Scr = serum creatinine (mg/dL), Scyst = serum cystatin C (mg/L)

The changes from reference in serum creatinine, eGFRcr<sub>CG</sub> and eGFRcr<sub>CKD-EPI</sub> and eGFRcyst<sub>CKD-EPI</sub> at Week 96 will be summarized by treatment arm and using descriptive statistics.

Within-treatment arm comparison versus reference at Week 96 will be assessed using Wilcoxon signed-rank test.

Stages of GFR at reference versus the minimum post-reference GFR value and the last available value will be summarized by count and percent of subjects. Kidney disease stages are defined as follows: 1 (Normal): GFR  $\geq$  90; 2 (Mild): GFR 60-89; 3 (Moderate): GFR 30-59; 4 (Severe): GFR 15-29; 5 (Renal Failure): GFR <15 mL/min).

In addition to the above, the number and proportion of subjects with a >25%, >50% and >75% decrease from reference will be tabulated.

#### 5.5.3.2. Proximal renal tubular function

### **Proteinuria by Quantitative Assessment**

Total urine protein, total urine albumin, urine protein to creatinine ratio (UPCR) and urine albumin to creatinine ratio (UACR) will be summarized by treatment arm and visit using descriptive statistics. The number and proportion of subjects with UACR and UPCR results in the following categories at Week 96 will be tabulates:

- UACR: < 30, 30 to 300, >300 mg/g
- UPCR:  $< 200 \text{ mg/g versus} \ge 200 \text{ mg/g}$

Median (Q1, Q3) percent change from reference over time will be plotted by treatment group.

The evolution over time of total urine protein and total urine albumin will also be presented.

### **Proteinuria by Urinalysis (Dipstick)**

Treatment-emergent proteinuria by urinalysis (dipstick) through Week 96 will be summarized by treatment group. Cross-tabulation of grades at Week 96 versus reference will also be presented.

#### **Other Renal Biomarkers**

Selected renal biomarkers retinol binding protein (RBP) and beta-2-microglobulin, RBP to creatinine ratio and beta-2-microglobulin to creatinine ratio will be summarized by treatment arm and visit using descriptive statistics.

The proportions of subjects with beta-2-microglobulin to creatinine ratio  $\leq 300 \,\mu\text{g/g}$  and  $\geq 300 \,\text{mg/g}$  will be tabulated.

The number and proportion of subjects with retinal binding protein to creatinine ratio results in the following categories at Week 96 will be tabulated:

- < 50 years of age (at the time of lab assessment): < 130 mcg/g creatinine,  $\geq$  130 mcg/g creatinine
- $\geq$  50 years of age (at the time of lab assessment): < 172 mcg/g creatinine,  $\geq$  172 mcg/g creatinine

### **Phosphate excretion**

Other renal biomarkers include urine fractional excretion of phosphate (FEPO4) that will be summarized by treatment arm and visit using descriptive statistics.

Urine fractional excretion of Phosphate (FEPO4) will be calculated as follows:

• Based on <u>unadjusted</u> serum creatinine: FEPO4 (%) = (SCr × UPO4) / (SPO4 × UCr) × 100 (%)

The reference, post-reference, and change from reference in FEPO4 will be summarized by treatment arm and visit using descriptive statistics. Median (Q1, Q3) change from baseline in FEPO4 over time will be plotted by treatment group.

# Subclinical renal proximal tubulopathy

Potential Markers of Renal Proximal Tubulopathy are

- 1. Increase in serum creatinine  $\geq 0.40$  mg/dL from reference.
- 2. Confirmed  $\geq$  2 grade level increase from reference in graded proteinuria
- 3. Confirmed  $\geq 1$  grade level increase from reference in graded hypophosphatemia
- 4. Confirmed ≥ 1 grade level increase from reference in graded glycosuria concurrent with serum glucose <=100 mg/dL (normoglycemic glycosuria)

A confirmed laboratory abnormality is defined as an abnormality observed at 2 consecutive postreference measurements or an abnormality observed at 1 measurement followed by study drug discontinuation A subclinical renal proximal tubulopathy is defined as confirmed abnormalities in any 2 out of the 4 renal parameters (serum creatinine and one or more of the 3 other markers of tubular dysfunction).

### 5.6. Vital Signs and Physical Examination Findings

#### 5.6.1. Definitions

The following vital signs parameters will be analyzed:

- pulse (bpm)
- systolic blood pressure, SBP (mmHg)
- diastolic blood pressure, DBP (mmHg)
- weight (kg)

Pulse, DBP and SBP are classified in the following abnormality codes:

| | Pulse (bpm) | DBP (mmHg) | SBP (mmHg) |
|---|---|---|---|
| Abnormally low | ≤ 50 | ≤ 50 | ≤ 90 |
| Grade 1 or mild | - | > 90 - < 100 | > 140 - < 160 |
| Grade 2 or moderate | - | ≥ 100 <b>-</b> < 110 | $\geq 160 - < 180$ |
| Grade 3 or severe | - | ≥ 110 | ≥ 180 |
| Abnormally high | ≥ 120 | - | - |

In determining abnormalities, the following rules are applied:

- worst grades/abnormalities are determined over the whole observational period for each trial phase separately, including post-reference scheduled *and* unscheduled measurements of that phase.
- The abnormalities 'abnormally low' and 'abnormally high'/grades are considered equally important, i.e. if a subject has as well an abnormally low as an abnormally high or graded value post-reference, both abnormalities are shown in the tables. (This means that the sum of the percentages can be more than 100%).

#### **Definition treatment-emergent:**

An abnormality will be considered treatment-emergent in a particular phase if it is worse than the reference corresponding to this phase. If the reference is missing, the abnormality is always considered as treatment-emergent. A shift from 'abnormally low' at reference to 'abnormally high' or 'grade ...' post reference (or vice versa) is also treatment-emergent.

### 5.6.2. Analysis methods

Descriptive statistics for the actual values and changes from reference per timepoint will be presented. For weight, comparative treatment phase and extended treatment phase will be presented for Initial switch group as well as Late switch group.

Cross-tabulations for the worst abnormalities versus reference per vital signs test will be produced.

Abnormal physical examination (symptom-directed) findings will be listed.

### 5.7. Bone Investigations

### 5.7.1. Definitions

#### Bone formation markers:

- Serum total alkaline phosphatase (ALP)
- Serum type 1 procollagen N-terminal (P1NP)

### Bone resorption markers:

Urinary or serum collagen type 1 cross-linked C-telopeptide (CTX)

#### Other:

- parathyroid hormone (PTH)
- 25-hydroxy vitamin D (25-OH VitD)

### Bone mineral density (BMD)

DXA scan of spine and hip (data of other regions, e.g. femoral neck may also be analyzed if available):

- BMD values
- BMD T- and Z-scores

The BMD status will be derived based on T-scores using the following categories:

| | Osteoporosis | Osteopenia | Normal |
|---------|--------------|--------------|--------|
| T-score | < -2.5 | -2.5 to < -1 | ≥ -1 |

# 5.7.2. Analysis methods

#### **Bone Biomarkers:**

Descriptive statistics for the actual values, changes and percent changes from reference per time point will be presented for each bone biomarker.

#### **DXA scan:**

Descriptive statistics for the actual values, change and percent changes from reference per time point will be presented for BMD parameters (including T- and Z-scores).

Within-treatment arm comparison versus reference at Week 96 will be assessed using Wilcoxon signed-rank test. The proportions of subjects with at least 3% change (decrease and increase separately) from reference in BMD will be presented at Week 96. Percent change from reference will also be tabulated based on thresholds; 5% and 7%.

BMD status will be tabulated (n, %) separately per time point, based on the T-score categories. Crosstabulations for the BMD status at Week 96 versus reference will be produced.

### **REFERENCES**

- 1. Guidance for Industry. Antiretroviral Drugs Using Plasma HIV RNA Measurements Clinical Considerations for Accelerated and Traditional Approval. October 2002.
- 2. Wensing AM, Calvez V, Günthard HF, et al. 2017 update of the drug resistance mutations in HIV-1. Top Antivir Med Dec2016/Jan2017; 24(4):132-141
- Cockcroft DW, Gault MH. Prediction of creatinine clearance from serum creatinine. Nephron. 1976;16:31-41

Statistical Analysis Plan TMC114IFD3013 (Week 96)

# **ATTACHMENTS**

### ATTACHMENT 1: PREDEFINED MAJOR PROTOCOL DEVIATIONS-BASED ON THE CURRENT LIST

The predefined major protocol deviations of this study are described in the Protocol Deviation Criteria document. The deviations that are considered to have an (possible) impact on efficacy are a subset of the predefined major protocol deviations and are indicated with 'Yes' below (column 'Exclude from Per Protocol Analysis') and if such deviations are reported for a subject, the subject will be excluded from the PP analysis.

In addition to the table below, subjects with a baseline HIV-1 RNA value ≥50 copies/mL and subjects with treatment adherence <65% (Late Switch group will use worst adherence from baseline to switch and from switch to week 96) per derivation ii will also be excluded from the per-protocol analysis set.

| Sequence<br>No. | Description | Protocol Deviation coded term (DVDECOD) | Exclude from PP |
|---|---|---|---|
| 1 | The subject has not been treated with a stable ARV regimen consisting of a bPI (limited to DRV or ATV with rtv or COBI, or LPV with rtv) combined with FTC/TDF only for at least 6 consecutive months preceding the screening visit. | Entered but did not satisfy criteria | Yes |
| 2 | <ul> <li>During the 12 months preceding screening while on stable ART: <ul> <li>The subject did not have at least 1 plasma HIV-1 RNA measurement &lt;50 copies/mL (or HIV-1 RNA undetectable by a local HIV-1 RNA test) occurring between 12 and 2 months prior to the screening visit while on the stable ARV regimen</li> <li>The subject has a documented plasma HIV-1 RNA concentrations ≥200 copies/mL.</li> <li>The subject has documented more than 1 plasma HIV-1 RNA concentrations ≥50 copies/mL (or HIV-1 RNA detectable by a local</li> </ul> </li> </ul> | Entered but did not satisfy criteria | Yes |

# Statistical Analysis Plan TMC114IFD3013

| | | | or ium rivicir in bo |
|---|---|---|---|
| | HIV-1 RNA test) | | |
| | or - The subject has at least 1 single documented plasma HIV-1 RNA | | |
| | concentrations ≥50 copies/mL and <200 copies/mL <b>but</b> had no subsequent VL measurement <50 HIV-1 RNA copies/mL at the latest 2 months prior to screening | | |
| | or | | |
| | • At the screening visit has HIV-1 RNA ≥50 copies/mL. | | |
| 3 | The subject has a history of failure on DRV treatment or any of DRV RAMs (V11I, V32I, L33F, I47V, I50V, I54M, I54L, T74P, L76V, I84V, L89V) (if historical genotypes are available) | Entered but did not satisfy criteria | Yes |
| 4 | The subject uses disallowed concomitant therapy specified in the protocol | Entered but did not satisfy criteria | Yes |
| 5 | The subject has any known allergies to the excipients of the D/C/F/TAF tablet, but the subject was randomized. | Entered but did not satisfy criteria | Yes |

| 6 | The dose of Investigational treatment arm (D/C/F/TAF tablet) or the active control arm (maintain current regimen consisting of a bPI with FTC/TDF) was temporarily not according to protocol for more than 4 consecutive weeks. | Received wrong treatment or incorrect dose (missed dose or extra dose) | Based on >4<br>weeks period.<br>In that case<br>classified as<br>major and<br>excluded from<br>PP |
|---|---|---|---|
| 7 | The intake of Investigational treatment arm (D/C/F/TAF tablet) or the active control arm (maintain current regimen consisting of a bPI with FTC/TDF) was interrupted for toxicity reasons for more than 4 consecutive weeks. | Received wrong treatment or incorrect dose (missed dose or extra dose) | |
| 8 | The intake of Investigational treatment arm (D/C/F/TAF tablet) or the active control arm (maintain current regimen consisting of a bPI with FTC/TDF) was interrupted for non-toxicity reasons for more than 4 consecutive weeks, or cumulatively for more than 8 weeks. | Received wrong treatment or incorrect dose (missed dose or extra dose | |
| 9 | The subject takes disallowed medication as defined per protocol. | Received a disallowed concomitant treatment | Yes (adjudication based on drug/class and duration). |
| 10 | The subject missed two or more consecutive planned visits in the trial | Other | Yes |
| 11 | Misallocation of Medkits was observed during Dosage and administration of study drug and subject treated differently than what they were randomized to for more than 4 weeks | Other | Yes |
| 12 | After achieving HIV-1 RNA <50 copies/mL, a single HIV-1 RNA value was ≥50 copies/mL, but a viral load retest or scheduled viral load test within 6 weeks of the previous VL result of ≥50 copies/mL was not collected (except for screening and baseline results) | Other | Yes |
| 13 | Subject missed the Week 96 visit. | Other | Yes |

<sup>\*</sup>Some sites assumed that protocol language "abnormal lab values that would lead to exclusion could be repeated once" applied also to viral load >50c/mL at screening.

\*\* Including subjects whose HIV-1 RNA was ≥50 copies/mL at screening, but had a HIV-1 RNA <50 copies/mL at a not per protocol defined retest during the screening period and who were randomized based on the latter HIV-1 RNA.

### **ATTACHMENT 2**

# **Adverse Events of Interest: List of Preferred Terms**

# **AEOI**

# **AEDECOD (MedDRA v20.0)**

| Rash AEOI | Acrodynia, Drug Eruption, Generalised erythema, Lupus miliaris disseminatus facei, Mucocutaneous rash, Rash, Rash erythematous, Rash generalised, Rash macular, Rash maculo-papular, Rash maculovesicular, Rash morbiliform, Rash papular, Rash pruritic, Rash rubelliform, Rash scarlatiniform, Red man syndrome, Rash vesicular, Rash follicular, Rash papulosquamous, Dermatitis, Dermatitis acneiform, Dermatitis allergic, Dermatitis herpetiformis, Skin necrosis, Skin reaction |
|---|---|
| Liver AEOI/Cholestasis and jaundice of hepatic origin | Bilirubin excretion disorder, Cholaemia, Cholestasis, Cholestatic liver injury, Cholestatic pruritus, Drug-induced liver injury, Hepatitis cholestatic, Hyperbilirubinaemia, Icterus index increased, Jaundice, Jaundice cholestatic, Jaundice hepatocellular, Mixed liver injury, Ocular icterus, Parenteral nutrition associated liver disease, Deficiency of bile secretion, Yellow skin |
Liver AEOI/Hepatic failure, fibrosis and cirrhosis and other liver damage related conditions

Acute hepatic failure, Acute on chronic liver failure, Acute yellow liver atrophy, Ascites, Asterixis, Bacterascites, Biliary cirrhosis, Biliary cirrhosis primary, Biliary fibrosis, Cholestatic liver injury, Chronic hepatic failure, Coma hepatic, Cryptogenic cirrhosis, Diabetic hepatopathy, Drug-induced liver injury, Duodenal varices, Gallbladder varices, Gastric variceal injection, Gastric variceal ligation, Gastric varices, Gastric varices haemorrhage, Hepatectomy, Hepatic atrophy, Hepatic calcification, Hepatic cirrhosis, Hepatic encephalopathy, Hepatic encephalopathy prophylaxis, Hepatic failure, Hepatic fibrosis, Hepatic hydrothorax, Hepatic infiltration eosinophilic, Hepatic lesion, Hepatic necrosis, Hepatic steato-fibrosis, Hepatic steatosis, Hepatitis fulminant, Hepatobiliary disease, Hepatocellular foamy cell syndrome, Hepatocellular injury, Hepatopulmonary syndrome, Hepatorenal failure, Hepatorenal syndrome, Hepatotoxicity, Intestinal varices, Liver and small intestine transplant, Liver and small intestine transplant, Liver dialysis, Liver disorder, Liver injury, Liver operation, Liver transplant, Lupoid hepatic cirrhosis, Minimal hepatic encephalopathy, Mixed liver injury, Nodular regenerative hyperplasia, Non-alcoholic fatty liver, Nonalcoholic steatohepatitis, Non-cirrhotic portal hypertension, Oedema due to hepatic disease, Oesophageal varices haemorrhage, Peripancreatic varices, Portal fibrosis, Portal hypertension, Portal hypertensive enteropathy, Portal hypertensive gastropathy, Portal vein cavernous transformation, Portal vein dilatation, Portopulmonary hypertension, Renal and liver transplant, Retrograde portal vein flow, Reye's syndrome, Reynold's syndrome, Splenic varices, Splenic varices haemorrhage, Steatohepatitis, Subacute hepatic failure, Varices oesophageal, Varicose veins of abdominal wall, Anorectal varices, Anorectal varices haemorrhage, Intrahepatic portal hepatic venous fistula, Peritoneovenous shunt, Portal shunt, Portal shunt procedure, Smallfor-size liver syndrome, Spider naevus, Splenorenal shunt, Splenorenal shunt procedure, Spontaneous intrahepatic portosystemic venous shunt, Stomal varices, Portal triaditis

Bromosulphthalein test abnormal, Child-Pugh-Turcotte score abnormal, Child-Pugh-Turcotte score increased, Computerised tomogram liver, Foetor hepaticus, Galactose elimination capacity test abnormal, Galactose elimination capacity test decreased, Gamma-glutamyltransferase abnormal, Gamma-glutamyltransferase increased, Guanase increased, Hepaplastin abnormal, Hepaplastin decreased, Hepatic artery flow decreased, Hepatic congestion, Hepatic enzyme abnormal, Hepatic enzyme decreased, Hepatic enzyme increased, Hepatic function abnormal, Hepatic hydrothorax, Hepatic hypertrophy, Hepatic mass, Hepatic pain, Hepatic sequestration, Hepatic vascular resistance increased, Hepatobiliary scan abnormal, Hepatomegaly, Hepatosplenomegaly, Hyperammonaemia, Hyperbilirubinaemia, Hypercholia, Hypertransaminasaemia, Kayser-Fleischer ring, Liver function test abnormal, Liver induration, Liver palpable, Liver scan abnormal, Liver tenderness, Mitochondrial aspartate aminotransferase increased, Molar ratio of total branched-chain amino acid to tyrosine, Oedema due to hepatic disease, Perihepatic discomfort, Retrograde portal vein flow, Total bile acids increased, Transaminases abnormal, Transaminases increased, Ultrasound liver abnormal, Urine bilirubin increased, X-ray hepatobiliary abnormal, 5'nucleotidase increased, Blood alkaline phosphatase abnormal, Blood alkaline phosphatase increased, Blood cholinesterase abnormal, Blood cholinesterase decreased, Deficiency of bile secretion, Glutamate dehydrogenase increased, Haemorrhagic ascites, Hepatic fibrosis marker abnormal, Hepatic fibrosis marker increased, Hypoalbuminaemia, Leucine

aminopeptidase increased, Liver function test decreased, Liver function test increased, Liver iron concentration abnormal, Liver iron concentration increased, Model for end stage liver disease score abnormal, Model for end stage liver disease score increased, Periportal oedema, Peritoneal fluid protein abnormal, Peritoneal fluid protein decreased, Peritoneal fluid protein increased, Pneumobilia, Portal vein flow decreased, Portal vein pressure increased, Retinol binding protein decreased, Urobilinogen urine

decreased, Urobilinogen urine increased, Liver palpable subcostal

Alanine aminotransferase abnormal, Alanine aminotransferase increased,

Ammonia abnormal, Ammonia increased, Ascites, Aspartate aminotransferase abnormal, Aspartate aminotransferase increased, Bacterascites, Bile output abnormal, Bile output decreased, Biliary ascites, Bilirubin conjugated abnormal, Bilirubin conjugated increased, Bilirubin urine present, Biopsy liver abnormal, Blood bilirubin abnormal, Blood

bilirubin increased, Blood bilirubin unconjugated increased,

Liver AEOI / Liver-related investigations, signs and symptoms

Liver AEOI / Hepatitis, non infectious

Acute graft versus host disease in liver, Allergic hepatitis, Autoimmune hepatitis, Chronic graft versus host disease in liver, Chronic hepatitis, Graft versus host disease in liver, Hepatitis, Hepatitis acute, Hepatitis cholestatic, Hepatitis chronic active, Hepatitis chronic persistent, Hepatitis fulminant, Hepatitis toxic, Ischaemic hepatitis, Lupus hepatitis, Non-alcoholic steatohepatitis, Radiation hepatitis, Steatohepatitis, Granulomatous liver disease, Liver sarcoidosis, Portal tract inflammation

Hyperglycaemia AEOI

Acquired lipoatrophic diabetes, Blood 1,5-anhydroglucitol decreased, Blood glucose increased, Diabetes complicating pregnancy, Diabetes mellitus, Diabetes mellitus inadequate control, Diabetes with hyperosmolarity, Diabetic arteritis, Diabetic coma, Diabetic hepatopathy, Diabetic hyperglycaemic coma, Diabetic hyperosmolar coma, Diabetic ketoacidosis, Diabetic ketoacidotic hyperglycaemic coma, Diabetic metabolic decompensation, Fructosamine increased, Fulminant type 1 diabetes mellitus, Gestational diabetes, Glucose tolerance impaired, Glucose tolerance impaired in pregnancy, Glucose urine present, Glycosuria, Glycosuria during pregnancy, Glycosylated haemoglobin increased, Hyperglycaemia, Hyperglycaemic seizure, Hyperglycaemic unconsciousness, Hyperosmolar hyperglycaemic state, Impaired fasting glucose, Insulin resistance, Insulin resistance syndrome, Insulin resistant diabetes, Insulinrequiring type 2 diabetes mellitus, Ketoacidosis, Ketonuria, Ketosis, Latent autoimmune diabetes in adults, Metabolic syndrome, Monogenic diabetes, Neonatal diabetes mellitus, Pancreatogenous diabetes, Type 1 diabetes mellitus, Type 2 diabetes mellitus, Type 3 diabetes mellitus, Urine ketone body present, Hyperglycaemic hyperosmolar nonketotic syndrome

Dyslipidaemia AEOI

Acquired lipoatrophic diabetes, Acquired mixed hyperlipidaemia, Apolipoprotein B/Apolipoprotein A-1 ratio increased, Autoimmune hyperlipidaemia, Blood cholesterol abnormal, Blood cholesterol decreased, Blood cholesterol esterase increased, Blood cholesterol increased, Blood triglycerides abnormal, Blood triglycerides decreased, Blood triglycerides increased, Diabetic dyslipidaemia, Dyslipidaemia, Familial hypertriglyceridaemia, Fat overload syndrome, High density lipoprotein abnormal, High density lipoprotein decreased, High density lipoprotein increased, Hypercholesterolaemia, Hyperlipidaemia, Hypertriglyceridaemia, Hypo HDL cholesterolaemia, Hypotriglyceridaemia, Intermediate density lipoprotein decreased, Intermediate density lipoprotein increased, LDL/HDL ratio decreased, LDL/HDL ratio increased, Lecithin-cholesterol acyltransferase deficiency, Lipid metabolism disorder, Lipids abnormal, Lipids decreased, Lipids increased, Lipoprotein (a) abnormal, Lipoprotein (a) decreased, Lipoprotein (a) increased, Low density lipoprotein abnormal, Low density lipoprotein decreased, Low density lipoprotein increased, Non-highdensity lipoprotein cholesterol decreased, Non-high-density lipoprotein cholesterol increased, Primary hypercholesterolaemia, Remnant hyperlipidaemia, Remnant-like lipoprotein particles increased, Total cholesterol/HDL ratio abnormal, Total cholesterol/HDL ratio decreased, Total cholesterol/HDL ratio increased, Type I hyperlipidaemia, Type II hyperlipidaemia, Type IIa hyperlipidaemia, Type IIb hyperlipidaemia, Type III hyperlipidaemia, Type IV hyperlipidaemia, Type V hyperlipidaemia, Very low density lipoprotein abnormal, Very low density lipoprotein decreased, Very low density lipoprotein increased

Lipodystrophy AEOI

Body fat disorder, Facial wasting, Fat redistribution, Fat tissue decreased, HIV lipodystrophy, Lipodystrophy acquired, Lipohypertrophy, Partial lipodystrophy

Immune reconstitution inflammatory AEOI

Immune reconstitution syndrome, Mycobacterium avium complex immune restoration disease, Immune Reconstitution Inflammatory Syndrome associated tuberculosis, Immune Reconstitution Inflammatory Syndrome associated Kaposi's sarcoma,

infarction, Myocardial necrosis, Myocardial reperfusion injury, Myocardial stunning, Papillary muscle infarction, Post procedural myocardial infarction, Postinfarction angina, Silent myocardial infarction, Troponin I increased, Troponin increased, Troponin T increased, Blood creatine phosphokinase abnormal, Blood creatine phosphokinase increased, Cardiac ventricular scarring, ECG electrically inactive area, ECG signs of myocardial infarction, Electrocardiogram Q wave abnormal, Electrocardiogram ST segment abnormal, Electrocardiogram ST segment elevation, Electrocardiogram ST-T segment elevation, Infarction, Myocardial necrosis marker increased, Scan myocardial perfusion abnormal, Vascular graft occlusion, Vascular stent occlusion, Vascular stent thrombosis, Angina pectoris, Angina unstable, Anginal equivalent, Arteriosclerosis coronary artery, Arteriospasm coronary, Coronary angioplasty, Coronary arterial stent insertion, Coronary artery bypass, Coronary artery disease, Coronary artery dissection, Coronary artery insufficiency, Coronary artery restenosis, Coronary artery stenosis, Coronary brachytherapy, Coronary bypass stenosis, Coronary endarterectomy, Coronary no-reflow phenomenon, Coronary ostial stenosis, Coronary revascularisation, Coronary vascular graft stenosis, Dissecting coronary artery aneurysm, ECG signs of myocardial ischaemia, External counterpulsation, Haemorrhage coronary artery, Ischaemic cardiomyopathy, Ischaemic mitral regurgitation, Microvascular coronary artery disease, Myocardial ischaemia, Percutaneous coronary intervention, Prinzmetal angina, Stress cardiomyopathy, Subclavian coronary steal syndrome, Subendocardial ischaemia, Arteriogram coronary abnormal, Cardiac stress test abnormal, Computerised tomogram coronary artery abnormal, Computerised tomogram coronary artery abnormal, Electrocardiogram ST

segment depression, Electrocardiogram ST-T segment abnormal, Electrocardiogram ST-T segment depression, Electrocardiogram T wave abnormal, Electrocardiogram T wave inversion, Exercise electrocardiogram abnormal, Exercise test abnormal, Post angioplasty restenosis, Stress echocardiogram abnormal, Vascular stent restenosis, Vascular stent

stenosis, Cardiac enzymes increased

Acute coronary syndrome, Acute myocardial infarction, Angina unstable, Blood creatine phosphokinase MB abnormal, Blood creatine phosphokinase MB increased, Coronary artery embolism, Coronary artery occlusion, Coronary artery reocclusion, Coronary artery thrombosis, Coronary bypass thrombosis, Coronary vascular graft occlusion, Kounis syndrome, Myocardial

Coronary artery AEOI

Severe skin AEOI

Acute generalised exanthematous pustulosis, Cutaneous vasculitis, Dermatitis bullous, Dermatitis exfoliative, Dermatitis exfoliative generalised, Drug rash with eosinophilia and systemic symptoms, Epidermal necrosis, Erythema multiforme, Exfoliative rash, Oculomucocutaneous syndrome, Skin necrosis, Stevens-Johnson syndrome, Toxic epidermal necrolysis, Toxic skin eruption, Acquired epidermolysis bullosa, Blister, Blister rupture, Bullous impetigo, Conjunctivitis, Corneal exfoliation, Drug eruption, Epidermolysis, Epidermolysis bullosa, Fixed drug eruption, Genital ulceration, HLA-B\*1502 assay positive, HLA-B\*5801 assay positive, Hypopharyngeal synechiae, Lip exfoliation, Mouth ulceration, Mucocutaneous ulceration, Mucosa vesicle, Mucosal erosion, Mucosal exfoliation, Mucosal necrosis, Mucosal ulceration, Nikolsky's sign, Noninfective conjunctivitis, Oral mucosal blistering, Oral mucosal exfoliation, Oral papule, Oropharyngeal blistering, Pemphigoid, Pemphigus, Penile exfoliation, Skin erosion, Skin exfoliation, Staphylococcal scalded skin syndrome, Stomatitis, Tongue exfoliation, Vaginal exfoliation, Vaginal ulceration, Vulval ulceration, Vulvovaginal rash, Vulvovaginal ulceration, Genital ulceration

Cardiac conduction AEOI/Conduction defects

Accessory cardiac pathway, Adams-Stokes syndrome, Agonal rhythm, Atrial conduction time prolongation, Atrioventricular block, Atrioventricular block complete, Atrioventricular block first degree, Atrioventricular block second degree, Atrioventricular conduction time shortened, Atrioventricular dissociation, Bifascicular block, Brugada syndrome, Bundle branch block, Bundle branch block bilateral, Bundle branch block left, Bundle branch block right, Conduction disorder, Defect conduction intraventricular, Electrocardiogram delta waves abnormal, Electrocardiogram PQ interval prolonged, Electrocardiogram PR prolongation, Electrocardiogram PR shortened, Electrocardiogram QRS complex prolonged, Electrocardiogram QT prolonged, Electrocardiogram repolarisation abnormality, Lenegre's disease, Long QT syndrome, Paroxysmal atrioventricular block, Sinoatrial block, Trifascicular block, Ventricular dyssynchrony, Wolff-Parkinson-White syndrome

Cardiac conduction AEOI / Torsade de pointes/QT prolongation

Electrocardiogram QT interval abnormal, Electrocardiogram QT prolonged, Long QT syndrome, Long QT syndrome congenital, Torsade de pointes, Ventricular tachycardia

Pancreas AEOI

Amylase abnormal, Hyperlipasaemia, Pancreatic enzymes abnormality, Amylase increased, Lipase abnormal, Pancreatic enzymes abnormal, Blood trypsine increased, Lipase increased, Pancreatic enzymes increased, Hyperamylasaemia, Lipase urine increased, Cullen's sign, Grey Turner's sign, Haemorrhagic necrotic pancreatitis, Hereditary pancreatitis, Ischaemic pancreatitis, Oedematous pancreatitis, Pancreatic abscess, Pancreatic haemorrhage, Pancreatic necrosis, Pancreatic phlegmon, Pancreatitis pseudocyst, Pancreatic pseudocyst drainage, Pancreatitis, Pancreatitis acute, Pancreatitis haemorrhagic, Pancreatitis necrotising, Pancreatitis relapsing, Pancreatorenal syndrome

Convulsions AEOI

Acquired epileptic aphasia, Acute encephalitis with refractory, repetitive partial seizures, Alcoholic seizure, Atonic seizures, Atypical benign partial epilepsy, Automatism epileptic, Autonomic seizure, Baltic myoclonic epilepsy, Benign familial neonatal convulsions, Benign rolandic epilepsy, Biotinidase deficiency, Change in seizure presentation, Clonic convulsion, Complex partial seizures, Convulsion in childhood, Convulsion neonatal, Convulsions local, Convulsive threshold lowered, Deja vu, Double cortex syndrome, Dreamy state, Drug withdrawal convulsions, Early infantile epileptic encephalopathy with burst-suppression, Eclampsia, Epilepsy, Epileptic aura, Epileptic psychosis, Febrile convulsion, Frontal lobe epilepsy, Generalised non-convulsive epilepsy, Generalised tonic-clonic seizure, Glucose transporter type 1 deficiency syndrome, Hemimegalencephaly, Hyperglycaemic seizure, Hypocalcaemic seizure, Hypoglycaemic seizure, Hyponatraemic seizure, Idiopathic generalised epilepsy, Infantile spasms, Juvenile myoclonic epilepsy, Lafora's myoclonic epilepsy, Lennox-Gastaut syndrome, Migraine-triggered seizure, Molybdenum cofactor deficiency, Myoclonic epilepsy, Myoclonic epilepsy and ragged-red fibres, Partial seizures, Partial seizures with secondary generalisation, Petit mal epilepsy, Polymicrogyria, Post stroke epilepsy, Post stroke seizure, Postictal headache, Postictal paralysis, Postictal psychosis, Postictal state, Post-traumatic epilepsy, Psychomotor seizures, Schizencephaly, Seizure, Seizure anoxic, Seizure cluster, Seizure like phenomena, Severe myoclonic epilepsy of infancy, Simple partial seizures, Status epilepticus, Sudden unexplained death in epilepsy, Temporal lobe epilepsy, Tonic clonic movements, Tonic convulsion, Tonic posturing, Topectomy, Uncinate fits, Convulsion, Grand mal convulsion

| Ocular AEOI (for Posterior Uveitis) | Acute zonal occult outer retinopathy, Anterior chamber cell, Anterior chamber fibrin, Anterior chamber flare, Anterior chamber inflammation, Aqueous fibrin, Autoimmune retinopathy, Autoimmune uveitis, Behcet's syndrome, Birdshot chorioretinopathy, Blau syndrome, Blindness, Blindness transient, Blindness unilateral, Chemical iritis, Chorioretinitis, Chorioretinopathy, Choroiditis, Ciliary hyperaemia, Cystoid macular oedema, Cytomegalovirus chorioretinitis, Eales' disease, Endophthalmitis, Exudative retinopathy, Eye inflammation, Fuchs' syndrome, Glaucomatocyclitic crises, Iridocyclitis, Iritis, Macular oedema, Non-infectious endophthalmitis, Noninfective chorioretinitis, Noninfective retinitis, Ocular toxicity, Ocular vasculitis, Optic discs blurred, Panophthalmitis, Photophobia, Photopsia, Retinal exudates, Retinal oedema, Retinal pigment epitheliopathy, Retinal toxicity, Retinal perivascular sheathing, Retinal vasculitis, Retinitis, Subretinal fluid, Sudden visual loss, Susac's syndrome, Sympathetic ophthalmia, Traumatic iritis, Tubulointerstitial nephritis and uveitis syndrome, Uveitis, Uveitis-glaucoma-hyphaema syndrome, Vision blurred, Visual acuity reduced, Visual field defect, Visual impairment, Vitreal cells, Vitreous floaters, Vitreous opacities, Vitritis, Vogt-Koyanagi-Harada syndrome |
|---|---|
| Renal AEOI (for PRT) / laboratory related events | Aminoaciduria, Beta-N-acetyl D glucosaminidase increased, Hyperphosphaturia, Renal glycosuria, Acquired aminoaciduria, Hyperchloraemia, Protein urine, Protein urine present, Proteinuria, Urine phosphorus abnormal, Beta-N-acetyl D glucosaminidase abnormal, Blood chloride increased, Blood phosphorus decreased, Blood potassium decreased, Blood uric acid abnormal, Blood uric acid decreased, Glucose urine present, Glycosuria, Hyperuricosuria, Hypokalaemia, Hypophosphataemia, Urine amino acid level abnormal, Urine amino acid level increased, Urine phosphorus increased, Urine uric acid abnormal, Urine uric acid increased |
| Renal AEOI (for PRT) / clinical events | Polydipsia, Polyuria, Nephropathy toxic, Renal tubular disorder, Chronic kidney disease, Fanconi syndrome, Fanconi syndrome acquired, Renal tubular acidosis |
| Bone AEOI (for fractures) /<br>Osteomalacia | Hypophosphataemic rickets, Osteomalacia, Renal osteodystrophy , Renal rickets, Rickets |
| Bone AEOI (for fractures) / Bone<br>Loss/atrophy | Bone atrophy, Bone decalcification, Bone density decreased, Bone formation decreased, Bone loss, Craniotabes, High turnover osteopathy, Hungry bone syndrome, Osteodystrophy, Osteolysis, Osteoporosis circumscripta cranii, Osteopenia, Senile osteoporosis, Osteoporosis, Cementoplasty |
| Bone AEOI (for fractures) / Fracture, possibly osteoporotic | Femoral neck fracture, Hip fracture, Lumbar vertebral fracture, Osteoporotic fracture, Spinal compression fracture, Spinal fracture, Thoracic vertebral fracture |

Bone AEOI (for fractures) / Fracture other

Acetabulum fracture, Ankle fracture, Atypical femur fracture, Atypical fracture, Avulsion fracture, Cervical vertebral fracture, Chance fracture, Clavicle fracture, Closed fracture manipulation, Comminuted fracture, Complicated fracture, Compression fracture, Elevation skull fracture, Epiphyseal fracture, External fixation of fracture, Femur fracture, Fibula fracture, Foot fracture, Forearm fracture, Fracture delayed union, Fracture displacement, Fracture malunion, Fracture nonunion, Fracture pain, Fracture reduction, Fracture treatment, Fracture treatments (excl skull and spine), Fractured ischium, Fractured sacrum, Fractured coccyx, Greenstick fracture, Hand fracture, Humerus fracture, Ilium fracture, Internal fixation of fracture, Limb fracture, Lower limb fracture, Multiple fractures, Open reduction of fracture, Open reduction of spinal fracture, Osteochondral fracture, Osteosynthesis, Patella fracture, Pathological fracture, Pelvic fracture, Periprosthetic fracture, Pubis fracture, Radius fracture, Rib fracture, Sacroiliac fracture, Scapula fracture, Skull fractured Skull fractured base, Spinal fusion fracture, Sternal fracture, Stress fracture, Tibia fracture, Torus fracture, Traumatic fracture, Ulna fracture, Upper limb fracture, Wrist fracture

Bone AEOI (for fractures) / Other Bone Events

Bone density abnormal, Bone disorder, Bone erosion, Bone lesion, Bone formation test abnormal, Bone fragmentation, Bone metabolism disorder, Bone pain, Bone resorption test abnormal, Bone scan abnormal, Bone development abnormal, Bone swelling, Epiphysiolysis, Nuclear magnetic resonance imaging spinal abnormal, Osteonecrosis, Osteonecrosis of jaw, Secondary sequestrum, Skeletal injury, Skeletal survey abnormal, Skull X-ray abnormal, Spinal X-ray abnormal, Vertebral lesion, Vertebral wedging, X-ray limb abnormal, X-ray of pelvis and hip abnormal, Bone densitometry

## **ATTACHMENT 3**

#### **ADR** grouped Terms

AE preferred terms (as available in AE Clinical database) are assigned an Adverse Drug Reaction System Organ Class (ADRSOC) and Adverse Drug Reaction (ADRCAT) according to the table below.

| Adverse Drug Reaction<br>System Organ Class | Adverse Drug Reaction | Adverse Event Preferred Term |
|---|---|---|
| GASTROINTESTINAL<br>DISORDERS | ABDOMINAL DISTENSION | ABDOMINAL DISTENSION |
| | ABDOMINAL PAIN | ABDOMINAL PAIN |
| | | ABDOMINAL PAIN LOWER |
| | | ABDOMINAL PAIN UPPER |
| | DIARRHOEA | DIARRHOEA |
| | | FREQUENT BOWEL MOVEMENTS |
| | DYSPEPSIA | DYSPEPSIA |
| | FLATULENCE | FLATULENCE |
| | NAUSEA | NAUSEA |
| | PANCREATITIS ACUTE | PANCREATITIS |
| | | PANCREATITIS ACUTE |
| | VOMITING | VOMITING |
| GENERAL DISORDERS<br>AND ADMINISTRATION<br>SITE CONDITIONS | ASTHENIA | ASTHENIA |
| | FATIGUE | FATIGUE |
| HEPATOBILIARY<br>DISORDERS | ACUTE HEPATITIS | HEPATITIS |
| | | HEPATITIS ACUTE |
| | | HEPATOTOXICITY |
| IMMUNE SYSTEM<br>DISORDERS | (DRUG) HYPERSENSITIVITY | DRUG HYPERSENSITIVITY |
| | | HYPERSENSITIVITY |
| | IMMUNE RECONSTITUTION SYNDROME | IMMUNE RECONSTITUTION INFLAMMATORY SYNDROME |
| | | IMMUNE RECONSTITUTION SYNDROME |
| METABOLISM AND<br>NUTRITION DISORDERS | ANOREXIA | DECREASED APPETITE |
| | DIABETES MELLITUS | DIABETES MELLITUS |
| | | DIABETES MELLITUS INADEQUATE CONTROL |
| | | TYPE 2 DIABETES MELLITUS |
| | | GLUCOSE TOLERANCE IMPAIRED |
| | LIPODYSTROPHY | FACIAL WASTING |

## Statistical Analysis Plan TMC114IFD3013

| FAT TISSUE INCREASED LUPOATROPHY MUSCULOSKELETAL AND CONNECTIVE TISSUE DISORDERS OSTEONECROSIS NERVOUS SYSTEM DISORDERS NERVOUS SYSTEM DISORDERS ABNORMAL DREAMS ANGIOEDEMA CIRCUMORAL CIRCUMORAL CONJUNCTIVAL OEDEMA CONJUNCTIVAL OEDEMA CORNEAL OEDEMA EYE OEDEMA EYE OEDEMA FACE OEDEMA FACE OEDEMA LUPOATROPM LARYNGEAL OEDEMA LARYN | | | Statistical Analysis Plan TMC1141FD3013 |
|---|---|---|---|
| LIPOATROPHY LIPOPYSTROPHY ACQUIRED LIPOPYSERTROPHY PARTIAL LIPOPYSTROPHY MUSCULOSKELETAL AND CONNECTIVE TISSUE DISORDERS OSTEONECROSIS OSTEONECROSIS OSTEONECROSIS OSTEONECROSIS OSTEONECROSIS OSTEONECROSIS OSTEONECROSIS NERVOUS SYSTEM DISORDERS ABNORMAL DREAMS ABNORMAL DREAMS BYPSYCHIATRIC DISORDERS REPRODUCTIVE SYSTEM AND BREAST DISORDERS ANGIOEDEMA ALLERGIC OEDEMA SUBCUTANEOUS TISSUE DISORDERS ANGIOEDEMA CORNEAL OEDEMA CONJUNCTIVAL OEDEMA EYE OEDEMA EYE OEDEMA EYE OEDEMA GINGIVAL OEDEMA GINGIVAL OEDEMA GINGIVAL OEDEMA LEYE OEDEMA LEYE OEDEMA LEYE OEDEMA LARYNGOTROME AGINGIVAL OEDEMA LARYNGOTROME AGINGIVAL OEDEMA LARYNGOTROME LARYNGOTROME ALARYNGOTROME ALARYNGOTRACHEAL OEDEMA LARYNGOTRACHEAL OEDEMA LIP SWELLING OCULORESPIRATORY SYNDROME OEDEMA MOUTH OROPHARYNGEAL SWELLING | | | FAT REDISTRIBUTION |
| LIPODYSTROPHY ACQUIRED LIPOHYPERTROPHY PARTIAL LIPODYSTROPHY MUSCULOSKELETAL AND CONNECTIVE TISSUE DISORDERS OSTEONECROSIS OSTEONECROSIS OSTEONECROSIS OSTEONECROSIS NERVOUS SYSTEM DISORDERS ABNORMAL DREAMS AND BREAST DISORDERS KIN AND BREAST DISORDERS ANGIOEDEMA ANGIOEDEMA ANGIOEDEMA CIRCUMORAL OEDEMA CONJUNCTIVAL OEDEMA EPIGLOTTIC OEDEMA EYE OEDEMA EYE SWELLING EYELID OEDEMA GINGIVAL OEDEMA GINGIVAL OEDEMA LIPODYSTROPHY GINGIVAL OEDEMA LARYNGOTRACHEAL OEDEMA LARYNGOTRACHEAL OEDEMA LARYNGOTRACHEAL OEDEMA LARYNGOTRACHEAL OEDEMA LIPODEMA LIPODEMA LIPODYSTROPHY MYALGIA MYALGIA MARGOTRACHEAL OEDEMA LIPODEMA OCULORESPIRATORY SYNDROME OEDEMA MOUTH OROPHARYNGEAL SWELLING | | | FAT TISSUE INCREASED |
| LIPOHYPERTROPHY PARTIAL LIPODYSTROPHY MUSCULOSKELETAL AND CONNECTIVE TISSUE DISORDERS OSTEONECROSIS OSTEONECROSIS OSTEONECROSIS NERVOUS SYSTEM DISORDERS NERVOUS SYSTEM DISORDERS ABNORMAL DREAMS AND BREAST DISORDERS SKIN AND SUBCUTANEOUS TISSUE DISORDERS ANGIOEDEMA ALLERGIC OEDEMA CONCUNCTIVAL CEDEMA CONCUNCTIVAL CEDEMA CONCULOTIVAL CEDEMA EYE GEDEMA EYE OEDEMA EYE SWELLING EYELID OEDEMA GINGIVAL OEDEMA GINGIVAL OEDEMA LIP CEDEMA LARYNGOTRACHEAL OEDEMA LIP OEDEMA LIP OEDEMA LIP OEDEMA OCOLURESPIRATORY SYNDROME OEDEMA MOUTH OROPHARYNGEAL SWELLING | | | LIPOATROPHY |
| PARTIAL LIPODYSTROPHY MYALGIA ABNORMAL DREAMS ABNORMAL DREAMS ABNORMAL DREAMS MYALGOMASTIA GYNAECOMASTIA MYPERTROPHY BREAST ALLERGIC OEDEMA ALLERGIC OEDEMA CIRCUMORAL OEDEMA CORNEAL OEDEMA EYE OEDEMA EYE OEDEMA EYE OEDEMA FACE OEDEMA FACE OEDEMA GINGIVAL OEDEMA GINGIVAL OEDEMA FACE OEDEMA LIPODYSTROPHY MYALGIA MYALGIA MYALGIA MYALGIA ABNORMAL DREAMS ALLERGIC OEDEMA CORLUMCTIVAL OEDEMA EYE OEDEMA EYE OEDEMA FACE OEDEMA FACE OEDEMA LARYNGOTA OEDEMA LARYNGOTA OEDEMA LARYNGOTA OEDEMA LIPOEDEMA LIPOEDEM | | | LIPODYSTROPHY ACQUIRED |
| MUSCULOSKELETAL AND CONNECTIVE TISSUE DISORDERS OSTEONECROSIS OSTEONECROSIS OSTEONECROSIS OSTEONECROSIS OSTEONECROSIS NERVOUS SYSTEM DISORDERS PSYCHIATRIC DISORDERS PSYCHIATRIC DISORDERS GYNAECOMASTIA ABNORMAL DREAMS ABNORMAL DRE | | | LIPOHYPERTROPHY |
| CONNECTIVE TISSUE DISORDERS OSTEONECROSIS OSTEONECROSIS OSTEONECROSIS NERVOUS SYSTEM DISORDERS ABNORMAL DREAMS REPRODUCTIVE SYSTEM AND BREAST DISORDERS ANGIOEDEMA ANGIOEDEMA ANGIOEDEMA ANGIOEDEMA ANGIOEDEMA ANGIOEDEMA CIRCUMORAL OEDEMA CORNEAL OEDEMA EYE OWEDEMA EYE OWEDEMA EYE OWEDEMA GIRGIVAL OEDEMA EYE OWEDEMA EYE OWEDEMA EYE OWEDEMA GIRGIVAL OEDEMA EYE OWEDEMA EYE OWEDEMA EYE OWEDEMA EYE OWEDEMA EYE OWEDEMA EYE OWEDEMA EYE SWELLING GIRGIVAL OEDEMA EYELID OEDEMA FACE OEDEMA LARYNGEAL OEDEMA LIP OEDEMA LIP OEDEMA LIP OEDEMA LIP OEDEMA OCULORESPIRATORY SYNDROME OEDEMA MOUTH OOROPHARYNGEAL SWELLING | | | PARTIAL LIPODYSTROPHY |
| NERVOUS SYSTEM DISORDERS PSYCHIATRIC DISORDERS PSYCHIATRIC ABNORMAL DREAMS ABNORMAL DREAMS SYNAECOMASTIA GYNAECOMASTIA HYPERTROPHY BREAST SKIN AND SUBCUTANEOUS TISSUE DISORDERS ANGIOEDEMA CORNIAL OEDEMA CORNIAL OEDEMA CORNIAL OEDEMA EYE OEDEMA GINGIVAL OEDEMA GINGIVAL OEDEMA GINGIVAL SWELLING GLEICH'S SYNDROME HEREDITARY ANGIOEDEMA LARYNGOTACHEAL OEDEMA LIP OEDEMA LIP OEDEMA LIP OEDEMA LIP OEDEMA LIP SWELLING LIP OEDEMA LIP SWELLING LIP OEDEMA LIP OEDEMA LIP OEDEMA LIP SWELLING LIP OEDEMA LIP SWELLING LIP OEDEMA LIP SWELLING LIP OEDEMA LIP SWELLING LIP OEDEMA LIP SWELLING OCULORESPIRATORY SYNDROME OCULORESPIRATORY SYNDROME OCULORESPIRATORY SYNDROME OCULORESPIRATORY SYNDROME OCULORESPIRATORY SYNDROME | CONNECTIVE TISSUE | MYALGIA | MYALGIA |
| DISORDERS PSYCHIATRIC DISORDERS REPRODUCTIVE SYSTEM AND BREAST DISORDERS SKIN AND SUBCUTANEOUS TISSUE DISORDERS ANGIOEDEMA ANGIOEDEMA ANGIOEDEMA ANGIOEDEMA ANGIOEDEMA ANGIOEDEMA ANGIOEDEMA CIRCUMORAL OEDEMA CONJUNCTIVAL OEDEMA EPIGLOTTIC OEDEMA EYE OEDEMA EYE SWELLING GINGIVAL OEDEMA GINGIVAL SWELLING GLEICH'S SYNDROME HEREDITARY ANGIOEDEMA LARYNGOTRACHEAL OEDEMA LIP SWELLING GCULORESPIRATORY SYNDROME LIP SWELLING LIP SWELLING LIP SWELLING LIP SWELLING LIP SWELLING OCULORESPIRATORY SYNDROME OEDEMA OCULORESPIRATORY SYNDROME OEDEMA OCULORESPIRATORY SYNDROME OEDEMA MOUTH OROPHARYNGEAL SWELLING | | OSTEONECROSIS | OSTEONECROSIS |
| DISORDERS REPRODUCTIVE SYSTEM AND BREAST DISORDERS SKIN AND BREAST DISORDERS SKIN AND SUBCUTANEOUS TISSUE DISORDERS ANGIOEDEMA ANGIOEDEMA ANGIOEDEMA CIRCUMORAL OEDEMA CONJUNCTIVAL OEDEMA CORNEAL OEDEMA EPIGLOTTIC OEDEMA EYE OEDEMA EYE OEDEMA EYE SWELLING EYELID OEDEMA GINGIVAL OEDEMA GINGIVAL OEDEMA LARYNGEAL OEDEMA LIP SWELLING OCULORESPIRATORY SYNDROME OEDEMA MOUTH OROPHARYNGEAL SWELLING | | HEADACHE | HEADACHE |
| AND BREAST DISORDERS HYPERTROPHY BREAST ALLERGIC OEDEMA ALLERGIC OEDEMA ALLERGIC OEDEMA ANGIOEDEMA ANGIOEDEMA CIRCUMORAL OEDEMA CONJUNCTIVAL OEDEMA CORNEAL OEDEMA EPIGLOTTIC OEDEMA EYE OEDEMA EYE SWELLING EYELID OEDEMA FACE OEDEMA GINGIVAL OEDEMA GINGIVAL OEDEMA LARYNGOEDEMA LARYNGOEDEMA LARYNGOEDEMA LARYNGOEDEMA LARYNGOEDEMA LIP OEDEMA LIP SWELLING OCULORESPIRATORY SYNDROME OEDEMA MOUTH OROPHARYNGEAL SWELLING | | ABNORMAL DREAMS | ABNORMAL DREAMS |
| SKIN AND SUBCUTANEOUS TISSUE DISORDERS ANGIOEDEMA ANGIOEDEMA CIRCUMORAL OEDEMA CONJUNCTIVAL OEDEMA CORNEAL OEDEMA EPIGLOTTIC OEDEMA EYE OEDEMA EYE SWELLING EYELID OEDEMA FACE OEDEMA GINGIVAL OEDEMA GINGIVAL OEDEMA GINGIVAL OEDEMA LARYNGEAL OEDEMA LARYNGEAL OEDEMA LARYNGEAL OEDEMA LARYNGOTRACHEAL OEDEMA LIP SWELLING OCULORESPIRATORY SYNDROME OEDEMA MOUTH OROPHARYNGEAL SWELLING | | GYNAECOMASTIA | GYNAECOMASTIA |
| SUBCUTANEOUS TISSUE DISORDERS ANGIOEDEMA CIRCUMORAL OEDEMA CONJUNCTIVAL OEDEMA CORNEAL OEDEMA EPIGLOTTIC OEDEMA EYE OEDEMA EYE SWELLING EYELID OEDEMA FACE OEDEMA GINGIVAL OEDEMA GINGIVAL OEDEMA LARYNGEAL OEDEMA LARYNGEAL OEDEMA LARYNGEAL OEDEMA LARYNGOTRACHEAL OEDEMA LIP OEDEMA LIP SWELLING OCULORESPIRATORY SYNDROME OEDEMA MOUTH OROPHARYNGEAL SWELLING | | | HYPERTROPHY BREAST |
| CIRCUMORAL OEDEMA CONJUNCTIVAL OEDEMA CORNEAL OEDEMA EPIGLOTTIC OEDEMA EPIGLOTTIC OEDEMA EYE OEDEMA EYE SWELLING EYELID OEDEMA FACE OEDEMA GINGIVAL OEDEMA GINGIVAL SWELLING GLEICH'S SYNDROME HEREDITARY ANGIOEDEMA LARYNGEAL OEDEMA LARYNGOTRACHEAL OEDEMA LIP OEDEMA LIP SWELLING OCULORESPIRATORY SYNDROME OEDEMA MOUTH OROPHARYNGEAL SWELLING | SUBCUTANEOUS TISSUE | ANGIOEDEMA | ALLERGIC OEDEMA |
| CONJUNCTIVAL OEDEMA CORNEAL OEDEMA EPIGLOTTIC OEDEMA EYE OEDEMA EYE SWELLING EYELID OEDEMA FACE OEDEMA GINGIVAL OEDEMA GINGIVAL SWELLING GLEICH'S SYNDROME HEREDITARY ANGIOEDEMA LARYNGEAL OEDEMA LARYNGEAL OEDEMA LIP OEDEMA LIP OEDEMA LIP SWELLING OCULORESPIRATORY SYNDROME OEDEMA MOUTH OROPHARYNGEAL SWELLING | | | ANGIOEDEMA |
| CONJUNCTIVAL OEDEMA CORNEAL OEDEMA EPIGLOTTIC OEDEMA EYE OEDEMA EYE SWELLING EYELID OEDEMA FACE OEDEMA GINGIVAL OEDEMA GINGIVAL SWELLING GLEICH'S SYNDROME HEREDITARY ANGIOEDEMA LARYNGEAL OEDEMA LARYNGEAL OEDEMA LIP OEDEMA LIP OEDEMA LIP SWELLING OCULORESPIRATORY SYNDROME OEDEMA MOUTH OROPHARYNGEAL SWELLING | | | |
| CORNEAL OEDEMA EPIGLOTTIC OEDEMA EYE OEDEMA EYE SWELLING EYELID OEDEMA FACE OEDEMA GINGIVAL OEDEMA GINGIVAL SWELLING GLEICH'S SYNDROME HEREDITARY ANGIOEDEMA LARYNGEAL OEDEMA LIP OEDEMA LIP SWELLING OCULORESPIRATORY SYNDROME OEDEMA MOUTH OROPHARYNGEAL SWELLING | | | CIRCUMORAL OEDEMA |
| EPIGLOTTIC OEDEMA EYE OEDEMA EYE SWELLING EYELID OEDEMA FACE OEDEMA GINGIVAL OEDEMA GINGIVAL SWELLING GLEICH'S SYNDROME HEREDITARY ANGIOEDEMA LARYNGEAL OEDEMA LIP OEDEMA LIP SWELLING OCULORESPIRATORY SYNDROME OEDEMA MOUTH OROPHARYNGEAL SWELLING | | | CONJUNCTIVAL OEDEMA |
| EYE OEDEMA EYE SWELLING EYELID OEDEMA FACE OEDEMA GINGIVAL OEDEMA GINGIVAL SWELLING GLEICH'S SYNDROME HEREDITARY ANGIOEDEMA LARYNGEAL OEDEMA LARYNGOTRACHEAL OEDEMA LIP OEDEMA LIP SWELLING OCULORESPIRATORY SYNDROME OEDEMA MOUTH OROPHARYNGEAL SWELLING | | | CORNEAL OEDEMA |
| EYE SWELLING EYELID OEDEMA FACE OEDEMA GINGIVAL OEDEMA GINGIVAL SWELLING GLEICH'S SYNDROME HEREDITARY ANGIOEDEMA LARYNGEAL OEDEMA LARYNGOTRACHEAL OEDEMA LIP OEDEMA LIP SWELLING OCULORESPIRATORY SYNDROME OEDEMA MOUTH OROPHARYNGEAL SWELLING | | | EPIGLOTTIC OEDEMA |
| EYELID OEDEMA FACE OEDEMA GINGIVAL OEDEMA GINGIVAL SWELLING GLEICH'S SYNDROME HEREDITARY ANGIOEDEMA LARYNGEAL OEDEMA LARYNGOTRACHEAL OEDEMA LIP OEDEMA LIP SWELLING OCULORESPIRATORY SYNDROME OEDEMA MOUTH OROPHARYNGEAL SWELLING | | | EYE OEDEMA |
| GINGIVAL OEDEMA GINGIVAL SWELLING GLEICH'S SYNDROME HEREDITARY ANGIOEDEMA LARYNGEAL OEDEMA LARYNGOTRACHEAL OEDEMA LIP OEDEMA LIP SWELLING OCULORESPIRATORY SYNDROME OEDEMA MOUTH OROPHARYNGEAL SWELLING | | | EYE SWELLING |
| GINGIVAL OEDEMA GINGIVAL SWELLING GLEICH'S SYNDROME HEREDITARY ANGIOEDEMA LARYNGEAL OEDEMA LARYNGOTRACHEAL OEDEMA LIP OEDEMA LIP SWELLING OCULORESPIRATORY SYNDROME OEDEMA MOUTH OROPHARYNGEAL SWELLING | | | EYELID OEDEMA |
| GINGIVAL SWELLING GLEICH'S SYNDROME HEREDITARY ANGIOEDEMA LARYNGEAL OEDEMA LARYNGOTRACHEAL OEDEMA LIP OEDEMA LIP SWELLING OCULORESPIRATORY SYNDROME OEDEMA MOUTH OROPHARYNGEAL SWELLING | | | FACE OEDEMA |
| GINGIVAL SWELLING GLEICH'S SYNDROME HEREDITARY ANGIOEDEMA LARYNGEAL OEDEMA LARYNGOTRACHEAL OEDEMA LIP OEDEMA LIP SWELLING OCULORESPIRATORY SYNDROME OEDEMA MOUTH OROPHARYNGEAL SWELLING | | | |
| GLEICH'S SYNDROME HEREDITARY ANGIOEDEMA LARYNGEAL OEDEMA LARYNGOTRACHEAL OEDEMA LIP OEDEMA LIP SWELLING OCULORESPIRATORY SYNDROME OEDEMA MOUTH OROPHARYNGEAL SWELLING | | | GINGIVAL OEDEMA |
| GLEICH'S SYNDROME HEREDITARY ANGIOEDEMA LARYNGEAL OEDEMA LARYNGOTRACHEAL OEDEMA LIP OEDEMA LIP SWELLING OCULORESPIRATORY SYNDROME OEDEMA MOUTH OROPHARYNGEAL SWELLING | | | GINGIVAL SWELLING |
| LARYNGEAL OEDEMA LARYNGOTRACHEAL OEDEMA LIP OEDEMA LIP SWELLING OCULORESPIRATORY SYNDROME OEDEMA MOUTH OROPHARYNGEAL SWELLING | | | |
| LARYNGEAL OEDEMA LARYNGOTRACHEAL OEDEMA LIP OEDEMA LIP SWELLING OCULORESPIRATORY SYNDROME OEDEMA MOUTH OROPHARYNGEAL SWELLING | | | HEREDITARY ANGIOEDEMA |
| LARYNGOTRACHEAL OEDEMA LIP OEDEMA LIP SWELLING OCULORESPIRATORY SYNDROME OEDEMA MOUTH OROPHARYNGEAL SWELLING | | | LARYNGEAL OEDEMA |
| LIP OEDEMA LIP SWELLING OCULORESPIRATORY SYNDROME OEDEMA MOUTH OROPHARYNGEAL SWELLING | | | LARYNGOTRACHEAL OEDEMA |
| LIP SWELLING OCULORESPIRATORY SYNDROME OEDEMA MOUTH OROPHARYNGEAL SWELLING | | | |
| OCULORESPIRATORY SYNDROME OEDEMA MOUTH OROPHARYNGEAL SWELLING | | | |
| OEDEMA MOUTH OROPHARYNGEAL SWELLING | | | |
| OROPHARYNGEAL SWELLING | | | |
| | | | PALATAL OEDEMA |

# D/C/F/TAF (darunavir/cobicistat/emtricitabine/tenofovir alafenamide)

# Statistical Analysis Plan TMC114IFD3013

| | | Statistical Analysis I fall Twic11411 D3013 |
|---|---|---|
| | | PERIORBITAL OEDEMA |
| | | PHARYNGEAL OEDEMA |
| | | SCLERAL OEDEMA |
| | | SMALL BOWEL ANGIOEDEMA |
| | | SWELLING FACE |
| | | SWOLLEN TONGUE |
| | | TONGUE OEDEMA |
| | | TRACHEAL OEDEMA |
| PRURI | ITUS | PRURIGO |
| | | PRURITUS |
| | | PRURITUS GENERALISED |
| RASH | | GENERALISED ERYTHEMA |
| | | RASH |
| | | RASH ERYTHEMATOUS |
| | | RASH GENERALISED |
| | | RASH MACULAR |
| | | RASH MACULO-PAPULAR |
| | | RASH MORBILLIFORM |
| | | RASH PAPULAR |
| | | RASH PRURITIC |
| STEVE | ENS-JOHNSON SYNDROME | STEVENS-JOHNSON SYNDROME |
| TOXIC | EPIDERMAL NECROLYSIS | TOXIC EPIDERMAL NECROLYSIS |
| URTIC | ARIA | URTICARIA |
| | | URTICARIA CHRONIC |
| | | URTICARIA PAPULAR |
| | | URTICARIA CHOLINERGIC |
| | | IDIOPATHIC URTICARIA |
| Acute ( | generalized exanthematous | Acute generalized exanthematous |
| pustulo | | pustulosis |
| Drug re | eaction with eosinophilia and | Drug reaction with eosinophilia and |
| system | nic symptoms | systemic symptoms |

#### **ATTACHMENT 4**

# List of AE Preferred Terms (MedDRAv 20.0) for Vital Signs Blood Pressure and Heart Rate

- Blood pressure abnormal
- Blood pressure decreased
- Blood pressure abnormal
- Blood pressure diastolic abnormal
- Blood pressure diastolic decreased
- Blood pressure diastolic increased
- Blood pressure increased
- Blood pressure systolic abnormal
- Blood pressure systolic decreased
- Blood pressure systolic increased
- Blood pressure abnormal
- Labile blood pressure
- Accelerated hypertenion
- Diastolic hypertension
- Essential hypertension
- Labile hypertension
- Malignant hypertension
- Systolic hypertension
- Diastolic hypotension
- Hypotension
- Heart rate abnormal
- Heart rate decreased
- Heart rate increased
- Heart rate irregular
- Bradycardia
- Tachycardia